CLINICAL TRIAL: NCT01459653
Title: International, Prospective, Open-label, Multicenter, Pharmacoepidemiological Study to Determine Predictors of Clinical Outcomes in Chemotherapy-treated Cancer Patients at Risk for Febrile Neutropenia and Treated Prophylactically With Filgrastim Biosimilar.
Brief Title: Multi-level Evaluation of Chemotherapy-induced Febrile Neutropenia Prophylaxis, Outcomes, and Determinants With Granulocyte-colony Stimulating Factor
Acronym: Monitor-GCSF
Status: Completed | Type: Observational
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Other Study IDs: EP06-502
Record Dates: First submitted 2011-08-30; First posted 2011-10-25 (Estimated); Results first posted 2015-07-07 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: Febrile Neutropenia; Cancer; Breast Cancer; Ovarian Cancer; Lung Cancer; Prostate Cancer; Multiple Myeloma; Bladder Cancer; B-cell Lymphoma
Keywords: Febrile neutropenia; cancer; chemotherapy,; primary prophylaxis; secondary prophylaxis; filgrastim; granulocyte colony stimulating factor; observational study; noninterventional study
MeSH Terms: conditions — Febrile Neutropenia; Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Multiple Myeloma; Urinary Bladder Neoplasms; Lymphoma, B-Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Only 1 group: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.

SUMMARY:
This international, prospective, observational, open-label, pharmaco-epidemiologic study observes cancer patients at risk for chemotherapy-induced febrile neutropenia (FN) who are receiving filgrastim biosimilar (EP2006) for primary or secondary FN prophylaxis to better describe the patient population at risk for FN and treated prophylactically in physician's best clinical judgement with filgrastim biosimilar (EP2006), to describe prophylaxis patterns involving filgrastim biosimilar (EP2006), and to evaluate hematology levels and variability in hematological outcomes, impact on chemotherapy delivery, radiotherapy, surgery, and mortality. Additionally the study aims to identify patient cohorts who are vulnerable to poor response to FN prophylaxis and experience break-through episodes of FN, understand the differences between prophylaxis responders and non-responders, and describe the degree to which prophylaxis of FN is in congruence with guideline recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults (age > / = 18 years)
* Diagnosed with one of the following types and stages of tumors: stage III or IV breast cancer; stage III or IV ovarian cancer; stage III or IV bladder cancer; stage III or IV lung cancer; metastatic prostate cancer; stage III or IV diffuse large B-cell lymphoma; multiple myeloma.
* Planned to receive primary prophylaxis with filgrastim biosimilar (EP2006) at the first cycle of chemotherapy (regardless of line of chemotherapy); or receiving secondary prophylaxis with filgrastim biosimilar (EP2006) irrespective of chemotherapy cycle.
* Treated with commercially available filgrastim biosimilar per physician's best clinical judgment and per current European filgrastim biosimilar (EP2006) label.
* Female patients must be either post-menopausal for one year or surgically sterile or using effective contraceptive methods such as barrier method with spermicide or an intra-uterine device. Oral contraceptive use is allowed.
* Informed written consent to participate in the study by patients or their legal guardian.

Exclusion Criteria:

* Patients with myeloid malignancies, with the exception of multiple myeloma.
* Sensitivity to filgrastim biosimilar or any other CSF.
* Hypersensitivity to E. coli-derived proteins.
* Radiotherapy to ≥ 20% of total body bone.
* Infection within two weeks of starting current line of chemotherapy.
* Patients with several medical condition(s) that in view of the investigator prohibits participation in the study.
* Patients with willfully negligent nonadherence to their cancer treatment.
* Use of any investigational agent in the 30 days prior to enrollment.
* Women of childbearing potential not using the contraception method(s) described above.
* Women who are breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar (EP2006) for primary or secondary prophylaxis for febrile neutropenia.
Sampling Method: Non-Probability Sample
Enrollment: 1496 (Actual)
Dates: Start 2010-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz GmBH, Study Chair — Sandoz GmbH
Locations (116):
- Austria (3):
  - Sandoz Investigational Site, Innsbruck
  - Sandoz Investigational Site, Kufstein
  - Sandoz Investigational Site, Leoben
- Belgium (2):
  - Sandoz Investigational Site, Deurne
  - Sandoz Investigational Site, Tournai
- Czechia (5):
  - Sandoz Investigational Site, Cheb
  - Sandoz Investigational Site, Chomutov
  - Sandoz Investigational Site, Prague
  - Sandoz Investigational Site, Teplice
  - Sandoz Investigational Site, Vítkovice
- France (31):
  - Sandoz Investigational Site, Agen
  - Sandoz Investigational Site, Arras
  - Sandoz Investigational Site, Avignon
  - Sandoz Investigational Site, Bayonne
  - Sandoz Investigational Site, Beauvais
  - Sandoz Investigational Site, Blois
  - Sandoz Investigational Site, Bois-Guillaume
  - Sandoz Investigational Site, Bordeaux
  - Sandoz Investigational Site, Boulogne-sur-Mer
  - Sandoz Investigational Site, Brest
  - Sandoz Investigational Site, Colmar
  - Sandoz Investigational Site, Compiègne
  - Sandoz Investigational Site, Gap
  - Sandoz Investigational Site, Grenoble
  - Sandoz Investigational Site, Libourne
  - Sandoz Investigational Site, Lille
  - Sandoz Investigational Site, Lyon
  - Sandoz Investigational Site, Marseille
  - Sandoz Investigational Site, Melun
  - Sandoz Investigational Site, Montauban
  - Sandoz Investigational Site, Montpellier
  - Sandoz Investigational Site, Nancy
  - Sandoz Investigational Site, Nîmes
  - Sandoz Investigational Site, Orléans
  - Sandoz Investigational Site, Paris
  - Sandoz Investigational Site, Perpignan
  - Sandoz Investigational Site, Pierre-Bénite
  - Sandoz Investigational Site, Poitiers
  - Sandoz Investigational Site, Reims
  - Sandoz Investigational Site, Sainte-Foy-lès-Lyon
  - Sandoz Investigational Site, Strasbourg
- Germany (21):
  - Sandoz Investigational Site, Berlin
  - Sandoz Investigational Site, Chemnitz
  - Sandoz Investigational Site, Coburg
  - Sandoz Investigational Site, Dortmund
  - Sandoz Investigational Site, Erlangen
  - Sandoz Investigational Site, Frankfurt
  - Sandoz Investigational Site, Gera
  - Sandoz Investigational Site, Hamburg
  - Sandoz Investigational Site, Heinsberg
  - Sandoz Investigational Site, Herne
  - Sandoz Investigational Site, Langen
  - Sandoz Investigational Site, Lehrte
  - Sandoz Investigational Site, Leipzig
  - Sandoz Investigational Site, Lübeck
  - Sandoz Investigational Site, Munich
  - Sandoz Investigational Site, Mülheim A. D. Ruhr
  - Sandoz Investigational Site, Weiden
  - Sandoz Investigational Site, Wismar
  - Sandoz Investigational Site, Witten
  - Sandoz Investigational Site, Wolfsburg
  - Sandoz Investigational Site, Würselen
- Hungary (6):
  - Sandoz Investigational Site, Budapest
  - Sandoz Investigational Site, Győr
  - Sandoz Investigational Site, Kecskemét
  - Sandoz Investigational Site, Pécs
  - Sandoz Investigational Site, Szekszárd
  - Sandoz Investigational Site, Szombathely
- Italy (19):
  - Sandoz Investigational Site, Avezzano
  - Sandoz Investigational Site, Avola
  - Sandoz Investigational Site, Bari
  - Sandoz Investigational Site, Campobasso
  - Sandoz Investigational Site, Colleferro
  - Sandoz Investigational Site, Cosenza
  - Sandoz Investigational Site, Cuneo
  - Sandoz Investigational Site, Frosinone
  - Sandoz Investigational Site, Gaeta
  - Sandoz Investigational Site, Genova
  - Sandoz Investigational Site, La Spezia
  - Sandoz Investigational Site, Matera
  - Sandoz Investigational Site, Milan
  - Sandoz Investigational Site, Monza
  - Sandoz Investigational Site, Rieti
  - Sandoz Investigational Site, Roma
  - Sandoz Investigational Site, S. Giovanni Rotondo
  - Sandoz Investigational Site, Sora
  - Sandoz Investigational Site, Torino
- Poland (9):
  - Sandoz Investigational Site, Bialystok
  - Sandoz Investigational Site, Brzozów
  - Sandoz Investigational Site, Bydgoszcz
  - Sandoz Investigational Site, Gdansk
  - Sandoz Investigational Site, Krakow
  - Sandoz Investigational Site, Lublin
  - Sandoz Investigational Site, Przemyśl
  - Sandoz Investigational Site, Warsaw
  - Sandoz Investigational Site, Wodzisław Śląski
- Romania (4):
  - Sandoz Investigational Site, Bucharest
  - Sandoz Investigational Site, Suceava
  - Sandoz Investigational Site, Târgu Mureş
  - Sandoz Investigational Site, Timișoara
- Spain (10):
  - Sandoz Investigational Site, Alicante
  - Sandoz Investigational Site, Barcelona
  - Sandoz Investigational Site, Benidorm Alicante
  - Sandoz Investigational Site, Bilbao
  - Sandoz Investigational Site, Donostia / San Sebastian
  - Sandoz Investigational Site, La Rioja
  - Sandoz Investigational Site, Lorca
  - Sandoz Investigational Site, Pamplona
  - Sandoz Investigational Site, Valencia
  - Sandoz Investigational Site, Vitoria-Gasteiz
- Switzerland (2):
  - Sandoz Investigational Site, Genolier
  - Sandoz Investigational Site, Zurich
- United Kingdom (4):
  - Sandoz Investigational Site, Cottingham
  - Sandoz Investigational Site, Liverpool
  - Sandoz Investigational Site, Rotherham
  - Sandoz Investigational Site, Scunthorpe

RESULTS

PARTICIPANT FLOW:
Groups:
- EP2006: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Period: Overall Study
Arm/Group | EP2006
Started | 1496
Completed | 828
Not Completed | 668

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are based on the evaluable sample, e.g. all patients who received at least one dose of the study medication, had no major protocol violation and have a minimum of enrollment cycle and either one follow-up cycle or study end data with valid outcome data (i.e., ANC or completed CIN/FN data).
Groups:
- EP2006, Evaluable Sample: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN. Only patients who had no major protocol violations and have a minimum of enrollment cycle and either one follow-up cycle or study end data with valid outcome data (i.e., ANC or completed CIN/FN data) belong to the evaluable sample and are analyzed.
Arm/Group | EP2006, Evaluable Sample
Number analyzed (Participants) | 1447
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 886
  Male | 561
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 1042
  African | 7
  Asian | 2
  Other | 1
  Missing | 395
Region of Enrollment [Number; unit: participants]
  France | 395
  Hungary | 143
  Czech Republic | 50
  Spain | 116
  Poland | 286
  Belgium | 3
  Romania | 64
  Austria | 27
  Germany | 145
  United Kingdom | 32
  Switzerland | 11
  Italy | 175
Height [Mean (Standard Deviation); unit: cm] — Number of participants analyzed: 1358
  cm | 165.6 (8.5)
Weight [Mean (Standard Deviation); unit: kg] — Number of participants analyzed: 1357
  kg | 72.1 (15.0)
Body-Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Number of participants analyzed: 1354
  kg/m^2 | 26.3 (5.0)
Medical history [Number; unit: participants] — Medical history for each patient was recorded. A patient can fall into more than one or none of the categories displayed.
  participants
    Bone pain | 116
    Joint pain | 78
    Muscle pain | 31
    Headache | 28
    Epistaxis | 8
    GI bleeding | 7
    Skin hemorrhage | 1
Comorbidities [Number; unit: participants] — Comorbidities for each patient were recorded. Only those comorbidities with a relative frequency of 5% or more are displayed in the table. A patient can fall into more than one or none of the categories displayed.
  participants
    Hypertension | 458
    Anemia | 138
    Diabetes Type II | 122
    Coronary disease | 93
    Allergies | 90
    COPD | 86
History of repeated infections [Number; unit: participants] — History of repeated infections for each patient was recoded. A patient can fall into more than one or none of the categories displayed.
  participants
    History of any repeated infection | 35
    Type of repeated infection (chronic) | 8
    Type of repeated infection (recurrent, acute) | 27
    1 infectious episode in past 3 months | 15
    2 infectious episodes in past 3 months | 7
    3 or more infectious episodes in past 3 months | 3
Cancer type [Number; unit: participants]
  Breast | 466
  Lung | 345
  Lymphoma (DLBCL) | 245
  Ovarian | 140
  Prostate | 102
  Multiple myeloma | 85
  Bladder | 64
Cancer stage & type [Number; unit: participants] — Table presents cancer stage by cancer stage. In addition, table presents cancer stage for all patients.
  participants
    Breast (stage III, n=466) | 267
    Breast (stage IV, n=466) | 194
    Lung (stage III, n=345) | 101
    Lung (stage IV, n=345) | 241
    Lymphoma (DLBCL) (stage III, n=245) | 103
    Lymphoma (DLBCL) (stage IV, n=245) | 135
    Ovarian (stage III, n=140) | 63
    Ovarian (stage IV, n=140) | 77
    Prostate (stage III, n=102) | 7
    Prostate (stage IV, n=102) | 95
    Multiple myeloma (stage III, n=85) | 53
    Multiple myeloma (stage IV, n=85) | 16
    Bladder (stage III, n=64) | 16
    Bladder (stage IV, n=64) | 48
    Overall, Stage III | 610
    Overall, Stage IV | 806
    Breast (unknown, n=466) | 5
    Lung (unknown, n=345) | 3
    Lymphoma (DLBCL) (unknown, n=245) | 7
    Multiple myeloma (unknown, N=85) | 16
    Overall, unknown | 31
Prior cancer treatments [Number; unit: participants] — Prior cancer treatments for all patients are recorded. A patient can have more than one prior cancer treatment. In addition, prior chemotherapy is also displayed by adjuvant or metastatic setting for those patients for whom this information was available.
  participants
    None | 518
    Surgery | 472
    Chemotherapy | 460
    Radiation therapy | 274
    Hormonal therapy | 198
    Targeted therapy | 45
    Bone marrow transplant | 12
    Other (including CAM) | 25
    Prior Chemotherapy, Adjuvant | 196
    Prior Chemotherapy, metastatic setting | 206
Cancer treatment [Number; unit: participants]
  Chemotherapy cycle at study entry (1) | 1046
  Chemotherapy cycle at study entry (2) | 221
  Chemotherapy cycle at study entry (3) | 93
  Chemotherapy cycle at study entry (4) | 44
  Chemotherapy cycle at study entry (5) | 26
  Chemotherapy cycle at study entry (6) | 17
History of prior CIN/FN and prior CIN/FN treatments [Number; unit: participants] — History of prior CIN/FN and prior CIN/FN treatment is recorded. A patient can fall into more than one or none of the categories displayed.
  participants
    Prior CIN grade 4 episodes (any) | 106
    Prior CIN grade 4 episodes (1) | 79
    Prior CIN grade 4 episodes (2) | 5
    Prior CIN grade 4 episodes (≥3) | 15
    Prior CIN grade 4 episodes (missing) | 7
    Prior FN | 27
    Hospitalization for CIN/FN | 33
    Any chemotherapy disturbance due to CIN/FN | 48
    Prior treatments for CIN/FN (CSF therapy) | 55
    Prior treatments for CIN/FN (antibiotics) | 44
    Prior treatments for CIN/FN (antiviral) | 0
    Prior treatments for CIN/FN (antifungal) | 7
    Prior treatments for CIN/FN (corticosteroids) | 5
    Prior treatments for CIN/FN (antipyretics) | 12
Treatment(s) for prior infections [Number; unit: participants] — 35 patients had prior infections. A patient can fall into more than category of prior infection treatment.
  participants
    Antibiotic | 33
    Antifungal | 2
    GCSF | 2
    Antiviral | 1
ECOG score at enrollment [Number; unit: participants] — ECOG (European Cooperative Oncology Group) score is a severity scale from 0 to 5 (highest) to grade toxicity and is defined as follows: 0=none, 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=lethal.
  ECOG is described in more detail by Oken et al, Am J Clin Oncol (CCT) 5:649-655, 1982.
  participants
    ECOG Score 0 | 553
    ECOG Score 1 | 652
    ECOG Score 2 | 121
    ECOG Score 3 | 26
    ECOG Score 4 | 1
    ECOG score Missing | 94
Cause(s) of prior repeated infections [Number; unit: participants] — 35 patients had prior repeated infections. Only those causes of prior repeated infections are shown with a frequency threshold of 5% based on the 35 patients with prior repeated infections are displayed. A patient may be counted in more than one or none of the categories displayed.
  participants
    Respiratory infections | 15
    Neutropenia | 11
    Cancer | 8
    High use of antibiotics | 3
    Urinary tract infections | 3
    Immunosuppression | 3
    Diabetes mellitus | 2
History of prior clinical events [Number; unit: participants] — Table shows number of patients with a specific prior clinical event. Only such events with a relative frequency threshold of 1% are displayed. A patient may be counted in more than one or none of the events displayed.
  participants
    Bone pain | 116
    Muscle pain | 31
    Joint pain | 78
    Headache | 28
Cancer stage by tumor type [Number; unit: participants] — DLBCL: Diffuse Large B-cell Lymphoma; Solid tumors include breast, lung, ovary, prostate and bladder; hematologic cancers include lymphoma (DLBCL) and multiple myeloma
  participants
    Solid tumor (n=1117), Stage III | 454
    Solid tumor (n=1117), Stage IV | 655
    Hematological tumor (n=330), Stage III | 156
    Hematological tumor (n=330), Stage IV | 151
    Solid tumor (n=1117), Stage unknown | 8
    Hematological tumor (n=330), Stage unknown | 23

OUTCOME MEASURES:

1. Primary Outcome: Chemotherapy Toxicity (%FN Risk)
Description: Objective 1: To describe the cancer patients requiring chemotherapy who, in their treating physician's best clinical judgment, are receiving EP2006 for the primary or secondary prophylaxis of FN in terms of demographics, clinical status, medical history, concomitant comorbid conditions and current status of disease, and prior and concomitant medications.
  Chemotherapy regimens were classified for FN risk (<10% risk, 10-20% risk or >20% risk) according to the published rates in the EORTC Guidelines under consideration of agent(s) and schedules.
  ANC=Absolute Neutrophil Count; CIN=Chemotherapy-Induced Neutropenia; FN=Febrile Neutropenia;
Time Frame: Enrollment cycle. Patients were evaluated at the enrollment cycle and then re-evaluated at each cycle for a maximum total of 6 cycles; however, the scheduling of these evaluations was left to the discretion of the physician.
Population: The evaluable sample includes all patients in the safety sample (all patients who received at least one dose of the study medication) who had no major protocol violation and have a minimum of enrollment cycle and either one follow-up cycle or study end data with valid outcome data. Please refer to baseline characteristics tables as well.
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1447
participants
  Low (<10%) | 154
  Medium (10-20%) | 650
  High (>20%) | 640
  Missing | 3

2. Primary Outcome: Cancer Treatment Type - Ever Received During Study
Description: Objective 1: To describe the cancer patients requiring chemotherapy who, in their treating physician's best clinical judgment, are receiving EP2006 for the primary or secondary prophylaxis of FN in terms of demographics, clinical status, medical history, concomitant comorbid conditions and current status of disease, and prior and concomitant medications.
  ANC=Absolute Neutrophil Count; CIN=Chemotherapy-Induced Neutropenia; FN=Febrile Neutropenia;
Time Frame: All cycles. Patients were evaluated at the enrollment cycle and then re-evaluated at each cycle for a maximum total of 6 cycles; however, the scheduling of these evaluations was left to the discretion of the physician, mean duration of study for 105 days
Population: The evaluable sample includes all patients in the safety sample (all patients who received at least one dose of the study medication) who had no major protocol violation and have a minimum of enrollment cycle and either one follow-up cycle or study end data with valid outcome data (i.e., ANC or completed CIN/FN data).
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1447
participants
  Surgery | 100
  Radiotherapy | 102
  Hormonal therapy | 85
  Targeted treatment | 89
  Bone marrow transplant | 31
  Other (e.g., CAM) | 98

3. Primary Outcome: Fever and Infections Ever During the Study
Description: as for outcome 2
Time Frame: as for outcome 2
Population: Evaluable consists of all patients who received at least one dose of study drug, who had no major protocol violations and have a minimum of enrollment cycle and either one follow-up cycle or study end data with valid outcome data (i.e. ANC or completed CIN/FN data).
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1447
participants
  Fever ever during study | 76
  Infections ever during study | 231

4. Primary Outcome: Clinical Events Ever During Study (Frequency Threshold: 5%)
Description: Objective 1: To describe the cancer patients requiring chemotherapy who, in their treating physician's best clinical judgment, are receiving EP2006 for the primary or secondary prophylaxis of FN in terms of demographics, clinical status, medical history, concomitant comorbid conditions and current status of disease, and prior and concomitant medications.
  ANC=Absolute Neutrophil Count; CIN=Chemotherapy-Induced Neutropenia; FN=Febrile Neutropenia
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1447
participants
  Bone pain | 357
  Thrombocytopenia | 230
  Serum LDH increase | 222
  Muscle pain | 210
  Joint pain | 200
  Serum GGT increase | 178
  Serum ALP increase | 168
  Other neurological symptoms | 102
  Headache | 100
  Blood uric acid increase | 88

5. Primary Outcome: Type of EP2006 Prophylaxis
Description: Objective 2: To describe EP2006 primary or secondary prophylaxis patterns for FN over up to 6 cycles of chemotherapy, with or without prior, concurrent, or later radiotherapy or surgery.
Time Frame: as for outcome 2
Population: Delayed Primary: EP2006 initiated in cycle 2 or later with no CIN/FN in prior cycle.
  True secondary: EP2006 initiated in cycle 2 or later following CIN/FN in prior cycle.
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1447
participants
  Primary (initiated in cycle1) | 1046
  Secondary (initiated in cycle2 or later) | 401
  Delayed primary | 245
  True secondary | 156

6. Primary Outcome: Type of EP2006 Prophylaxis by Gender
Description: as for outcome 5
Time Frame: as for outcome 2
Population: Evaluable sample by gender
Measure: Number; unit: participants
Groups:
- EP2006: Male: Male cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006: Female: Female cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Arm/Group | EP2006: Male | EP2006: Female
Number analyzed (Participants) | 561 | 886
participants
  Primary (initiated in cycle1) | 397 | 649
  Secondary (initiated in cycle2 or later) | 164 | 237
Statistical Analysis 1: Comparison: EP2006: Male vs EP2006: Female; Test type: Superiority or Other; p = 0.3038, Chi-squared; Odds Ratio (OR) = 0.8840, 95% CI 2-sided [0.6989 to 1.1182]

7. Primary Outcome: Type of EP 2006 Prophylaxis by Age Group
Description: as for outcome 5
Time Frame: as for outcome 2
Population: Evaluable sample by age
Measure: Number; unit: participants
Groups:
- EP2006: <65 Years: Cancer patients <65 years treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006: >=65 Years: Cancer patients >=65 years treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Arm/Group | EP2006: <65 Years | EP2006: >=65 Years
Number analyzed (Participants) | 849 | 598
participants
  Primary (initiated in cycle1) | 626 | 420
  Secondary, initiated in cycle2 or later | 223 | 178
Statistical Analysis 1: Comparison: EP2006: <65 Years vs EP2006: >=65 Years; Test type: Superiority or Other; p = 0.1432, Chi-squared; Odds Ratio (OR) = 1.1897, 95% CI 2-sided [0.9428 to 1.5012]

8. Primary Outcome: Type of EP 2006 Prophylaxis by Tumor Type
Description: as for outcome 5
Time Frame: as for outcome 2
Population: Evaluable sample by tumor type
Measure: Number; unit: participants
Groups:
- EP2006: Solid Tumor: Cancer patients with solid tumor treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006: Hematological Tumor: Cancer patients with hematological tumor treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Arm/Group | EP2006: Solid Tumor | EP2006: Hematological Tumor
Number analyzed (Participants) | 1117 | 330
participants
  Primary (initiated in cycle1) | 801 | 245
  Secondary (initiated in ≥cycle2) | 316 | 85
Statistical Analysis 1: Comparison: EP2006: Solid Tumor vs EP2006: Hematological Tumor; Test type: Superiority or Other; p = 0.6483, Chi-squared; Odds Ratio (OR) = 0.8794, 95% CI 2-sided [0.5063 to 1.5276]

9. Primary Outcome: Concomitant Antibiotic Prophylaxis
Description: as for outcome 5
Time Frame: as for outcome 2
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1447
participants
  Concomitant antibiotic prophylaxis | 175
  No Concomitant antibiotic prophylaxis | 1261
  Missing | 11

10. Primary Outcome: EP2006 Dose (All Cycles)
Description: as for outcome 5
Time Frame: as for outcome 2
Population: All cycles from patients in the evaluable sample
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1447
Number analyzed (cycles) | 5986
cycles
  30 MIU/day | 3182
  48 MIU/day | 2756
  Other | 48

11. Primary Outcome: EP2006 Dose (Enrollment Cycle)
Description: as for outcome 5
Time Frame: as for outcome 1
Population: Number of participants at enrollment cycle with dose data
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1434
participants
  30 MIU/day | 815
  48 MIU/day | 610
  Other | 9

12. Primary Outcome: EP2006 Dose (Cycle 1)
Description: as for outcome 5
Time Frame: Cycle 1. Patients were evaluated at the enrollment cycle and then re-evaluated at each cycle for a maximum total of 6 cycles; however, the scheduling of these evaluations was left to the discretion of the physician.
Population: Number of participants at cycle 1 with dose data
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1036
participants
  30 MIU/day | 593
  48 MIU/day | 434
  Other | 9

13. Primary Outcome: EP2006 Dose (Cycle 2)
Description: as for outcome 5
Time Frame: Cycle 2. Patients were evaluated at the enrollment cycle and then re-evaluated at each cycle for a maximum total of 6 cycles; however, the scheduling of these evaluations was left to the discretion of the physician.
Population: Number of participants at cycle 2 with dose data
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1143
participants
  30 MIU/day | 627
  48 MIU/day | 507
  Other | 9

14. Primary Outcome: EP2006 Dose (Cycle 3)
Description: as for outcome 5
Time Frame: Cycle 3. Patients were evaluated at the enrollment cycle and then re-evaluated at each cycle for a maximum total of 6 cycles; however, the scheduling of these evaluations was left to the discretion of the physician.
Population: Number of participants at cycle 3 with dose data
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1125
participants
  30 MIU/day | 597
  48 MIU/day | 519
  Other | 9

15. Primary Outcome: EP2006 Dose (Cycle 4)
Description: as for outcome 5
Time Frame: Cycle 4. Patients were evaluated at the enrollment cycle and then re-evaluated at each cycle for a maximum total of 6 cycles; however, the scheduling of these evaluations was left to the discretion of the physician.
Population: Number of participants at cycle 4 with dose data
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1045
participants
  30 MIU/day | 548
  48 MIU/day | 490
  Other | 7

16. Primary Outcome: EP2006 Dose (Cycle 5)
Description: as for outcome 5
Time Frame: Cycle 5. Patients were evaluated at the enrollment cycle and then re-evaluated at each cycle for a maximum total of 6 cycles; however, the scheduling of these evaluations was left to the discretion of the physician.
Population: Number of participants at cycle 5 with dose data
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 862
participants
  30 MIU/day | 431
  48 MIU/day | 424
  Other | 7

17. Primary Outcome: EP2006 Dose (Cycle 6)
Description: as for outcome 5
Time Frame: Cycle 6. Patients were evaluated at the enrollment cycle and then re-evaluated at each cycle for a maximum total of 6 cycles; however, the scheduling of these evaluations was left to the discretion of the physician.
Population: Number of participants at cycle 6 with dose data
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 775
participants
  30 MIU/day | 386
  48 MIU/day | 382
  Other | 7

18. Primary Outcome: EP2006 Dose by Patient Weight: Cycle Level
Description: as for outcome 5
Time Frame: as for outcome 2
Population: All cycles treated
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Groups:
- EP2006: <=65kg: Cancer patients weighing <=65kg treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006: >65kg: Cancer patients weighing >65kg treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Arm/Group | EP2006: <=65kg | EP2006: >65kg
Number analyzed (Participants) | 568 | 857
Number analyzed (cycles) | 2272 | 3666
cycles
  30 MIU/day | 1501 | 1681
  48 MIU/day | 771 | 1985
Statistical Analysis 1: Comparison: EP2006: <=65kg vs EP2006: >65kg; Test type: Superiority or Other; p < 0.0001, Chi-squared; Odds Ratio (OR) = 2.2989, 95% CI 2-sided [1.8113 to 2.9177]

19. Primary Outcome: EP2006 Dose by Tumor Type: Cycle Level
Description: as for outcome 5
Time Frame: as for outcome 2
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Arm/Group | EP2006: Solid Tumor | EP2006: Hematological Tumor
Number analyzed (Participants) | 1104 | 328
Number analyzed (cycles) | 4609 | 1329
cycles
  30 MIU/day | 2296 | 886
  48 MIU/day | 2313 | 443
Statistical Analysis 1: Comparison: EP2006: Solid Tumor vs EP2006: Hematological Tumor; Test type: Superiority or Other; p < 0.0001, Chi-squared; Odds Ratio (OR) = 0.4963, 95% CI 2-sided [0.3730 to 0.6605]

20. Primary Outcome: Patient Weight by Tumor Type (Solid Tumor vs. Hematological Tumor)
Description: as for outcome 5
Time Frame: as for outcome 2
Population: Evaluable sample by tumor type
Measure: Number; unit: participants
Arm/Group | EP2006: Solid Tumor | EP2006: Hematological Tumor
Number analyzed (Participants) | 1117 | 330
participants
  ≤65 kg | 441 | 135
  >65 kg | 676 | 195
Statistical Analysis 1: Comparison: EP2006: Solid Tumor vs EP2006: Hematological Tumor; Test type: Superiority or Other; p = 0.7509, Chi-squared; Odds Ratio (OR) = 0.9451, 95% CI 2-sided [0.6671 to 1.3391]

21. Primary Outcome: EP2006 Dose by Chemotherapy Toxicity: Cycle Level
Description: as for outcome 5
Time Frame: as for outcome 2
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Groups:
- EP2006: Risk <10%: Cancer patients with chemotherapy toxicity <10% treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006: Risk 10-20%: Cancer patients with chemotherapy toxicity 10-20% treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006: Risk >20%: Cancer patients with chemotherapy toxicity >20% treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Arm/Group | EP2006: Risk <10% | EP2006: Risk 10-20% | EP2006: Risk >20%
Number analyzed (Participants) | 151 | 647 | 631
Number analyzed (cycles) | 546 | 2534 | 2843
cycles
  30 MIU/day | 357 | 1375 | 1441
  48 MIU/day | 189 | 1159 | 1402
Statistical Analysis 1: Comparison: EP2006: Risk <10% vs EP2006: Risk 10-20% vs EP2006: Risk >20%; Test type: Superiority or Other; p = 0.0067, Chi-squared; Odds Ratio (OR) = 1.2683, 95% CI 2-sided [1.0680 to 1.5061]

22. Primary Outcome: EP2006 Day of Initiation: All Cycles
Description: as for outcome 5
Time Frame: as for outcome 2
Population: Cycles of patients in evaluable sample with day of initiation of study drug
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1447
Number analyzed (cycles) | 5930
days | 3.1 (3.0)

23. Primary Outcome: EP2006 Day of Initiation: Cycle 1
Description: as for outcome 5
Time Frame: as for outcome 12
Population: Cycles of patients in evaluable sample with study drug initiation day at cycle 1
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1017
Number analyzed (cycles) | 1017
days | 3.4 (3.2)

24. Primary Outcome: EP2006 Day of Initiation: Cycle 2
Description: as for outcome 5
Time Frame: as for outcome 13
Population: Cycles of patients in evaluable sample with study drug initiation day at cycle 2
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1132
Number analyzed (cycles) | 1132
days | 3.1 (3.0)

25. Primary Outcome: EP2006 Day of Initiation: Cycle 3
Description: as for outcome 5
Time Frame: as for outcome 14
Population: Cycles of patients in evaluable sample with study drug initiation day at cycle 3
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1111
Number analyzed (cycles) | 1111
days | 3.0 (2.9)

26. Primary Outcome: EP2006 Day of Initiation: Cycle 4
Description: as for outcome 5
Time Frame: as for outcome 15
Population: Cycles of patients in evaluable sample with study drug initiation day at cycle 4
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1038
Number analyzed (cycles) | 1038
days | 3.0 (2.9)

27. Primary Outcome: EP2006 Day of Initiation: Cycle 5
Description: as for outcome 5
Time Frame: as for outcome 16
Population: Cycles of patients in evaluable sample with study drug initiation day at cycle 5
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 858
Number analyzed (cycles) | 858
days | 2.9 (2.9)

28. Primary Outcome: EP2006 Day of Initiation: Cycle 6
Description: as for outcome 5
Time Frame: as for outcome 17
Population: Cycles of patients in evaluable sample with study drug initiation day at cycle 6
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 774
Number analyzed (cycles) | 774
days | 3.0 (2.9)

29. Primary Outcome: EP2006 Day of Initiation by Tumor Type (Solid Tumor vs. Hematological Tumor): Cycle Level
Description: as for outcome 5
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006: Solid Tumor | EP2006: Hematological Tumor
Number analyzed (Participants) | 1103 | 320
Number analyzed (cycles) | 4614 | 1316
days | 2.6 (2.7) | 4.8 (3.3)
Statistical Analysis 1: Comparison: EP2006: Solid Tumor vs EP2006: Hematological Tumor; Test type: Superiority or Other; p < 0.0001, ANOVA; degrees of freedom: 4507; Slope = 1.0628, 95% CI 2-sided [0.6382 to 1.4874]

30. Primary Outcome: EP2006 Day of Initiation by Prophylaxis Type: Cycle Level
Description: as for outcome 5
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Groups:
- EP2006: Primary Prophylaxis: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary prophylaxis for FN.
- EP2006: Secondary Prophylaxis: Cancer patients treated with chemotherapy as and who are prescribed commercially available filgrastim biosimilar for secondary prophylaxis for FN.
Arm/Group | EP2006: Primary Prophylaxis | EP2006: Secondary Prophylaxis
Number analyzed (Participants) | 1033 | 390
Number analyzed (cycles) | 4700 | 1230
days | 3.2 (3.0) | 2.6 (2.9)
Statistical Analysis 1: Comparison: EP2006: Primary Prophylaxis vs EP2006: Secondary Prophylaxis; Test type: Superiority or Other; p = 0.0103, ANOVA; degrees of freedom: 4507; Slope = -0.2739, 95% CI 2-sided [-0.4832 to -0.0646]

31. Primary Outcome: EP2006 Day of Initiation by Chemotherapy Toxicity: Cycle Level
Description: as for outcome 5
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Groups:
- EP2006: <10% Risk: Cancer patients treated with chemotherapy with low toxicity (<10% risk) and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006: 10-20% Risk: Cancer patients treated with chemotherapy with medium toxicity (10-20% risk) and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006: >20% Risk: Cancer patients treated with chemotherapy with high toxicity (>20% risk) and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Arm/Group | EP2006: <10% Risk | EP2006: 10-20% Risk | EP2006: >20% Risk
Number analyzed (Participants) | 150 | 637 | 633
Number analyzed (cycles) | 542 | 2504 | 2869
days | 2.3 (2.9) | 3.0 (3.0) | 3.3 (3.0)
Statistical Analysis 1: Comparison: EP2006: <10% Risk vs EP2006: 10-20% Risk vs EP2006: >20% Risk; Test type: Superiority or Other; p < 0.0001, ANOVA; degrees of freedom: 4495; Slope = 0.3812, 95% CI 2-sided [0.2330 to 0.5295]

32. Primary Outcome: EP2006 Treatment Duration in Any Cycle
Description: as for outcome 5
Time Frame: as for outcome 2
Population: All cycles from patients in the evaluable sample with study drug duration
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1426
Number analyzed (cycles) | 5942
days | 5.1 (2.3)

33. Primary Outcome: EP2006 Treatment Duration in Cycle 1
Description: as for outcome 5
Time Frame: as for outcome 12
Population: Cycles of participants in evaluable sample with study drug duration in cycle 1
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1025
Number analyzed (cycles) | 1025
days | 5.2 (2.2)

34. Primary Outcome: EP2006 Treatment Duration in Cycle 2
Description: as for outcome 5
Time Frame: as for outcome 13
Population: Cycles of participants in evaluable sample with study drug duration in cycle 2
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1134
Number analyzed (cycles) | 1134
days | 5.1 (2.3)

35. Primary Outcome: EP2006 Treatment Duration in Cycle 3
Description: as for outcome 5
Time Frame: as for outcome 14
Population: Cycles of participants in evaluable sample with study drug duration in cycle 3
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1117
Number analyzed (cycles) | 1117
days | 5.2 (2.3)

36. Primary Outcome: EP2006 Treatment Duration in Cycle 4
Description: as for outcome 5
Time Frame: as for outcome 15
Population: Cycles of participants in evaluable sample with study drug duration in cycle 4
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1039
Number analyzed (cycles) | 1039
days | 5.1 (2.3)

37. Primary Outcome: EP2006 Treatment Duration in Cycle 5
Description: as for outcome 5
Time Frame: as for outcome 16
Population: Cycles of participants in evaluable sample with study drug duration in cycle 5
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 856
Number analyzed (cycles) | 856
days | 5.1 (2.4)

38. Primary Outcome: EP2006 Treatment Duration in Cycle 6
Description: as for outcome 5
Time Frame: as for outcome 17
Population: Cycles of participants in evaluable sample with study drug duration in cycle 6
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 771
Number analyzed (cycles) | 771
days | 5.0 (2.4)

39. Primary Outcome: EP2006 Duration by Tumor Type: Cycle Level
Description: as for outcome 5
Time Frame: as for outcome 2
Population: Evaluable sample by tumor type with data
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006: Solid Tumor | EP2006: Hematological Tumor
Number analyzed (Participants) | 1103 | 323
Number analyzed (cycles) | 4619 | 1323
days | 5.14 (2.24) | 5.03 (2.56)
Statistical Analysis 1: Comparison: EP2006: Solid Tumor vs EP2006: Hematological Tumor; Test type: Superiority or Other; p = 0.0677, ANOVA; degrees of freedom: 4516; Slope = 0.1031, 95% CI 2-sided [-0.0075 to 0.2136]

40. Primary Outcome: EP2006 Duration by Prophylaxis Type: Cycle Level
Description: as for outcome 5
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Groups:
- EP2006: Secondary Prophylaxis: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for secondary prophylaxis for FN.
Arm/Group | EP2006: Primary Prophylaxis | EP2006: Secondary Prophylaxis
Number analyzed (Participants) | 1033 | 393
Number analyzed (cycles) | 4703 | 1239
days | 5.1 (2.2) | 5.2 (2.7)
Statistical Analysis 1: Comparison: EP2006: Primary Prophylaxis vs EP2006: Secondary Prophylaxis; Test type: Superiority or Other; p = 0.8968, ANOVA; degrees of freedom: 4516; Slope = 0.0018, 95% CI 2-sided [-0.0259 to 0.0295]

41. Primary Outcome: EP2006 Duration by Chemotherapy Toxicity: Cycle Level
Description: as for outcome 5
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: cycles
Arm/Group | EP2006: <10% Risk | EP2006: 10-20% Risk | EP2006: >20% Risk
Number analyzed (Participants) | 150 | 638 | 635
Number analyzed (cycles) | 541 | 2513 | 2875
days | 4.6 (2.4) | 5.0 (2.2) | 5.3 (2.4)
Statistical Analysis 1: Comparison: EP2006: <10% Risk vs EP2006: 10-20% Risk vs EP2006: >20% Risk; Test type: Superiority or Other; p < 0.0001, ANOVA; degrees of freedom: 4505; Slope = 0.0741, 95% CI 2-sided [-0.0452 to 0.1029]

42. Primary Outcome: Percentage of Patients With Each EORTC-identified Risk Factors for FN at Baseline
Description: Objective 3: To determine the extent to which the primary and secondary prophylaxis of FN in cancer patients is in congruence with the EORTC best practice guidelines and dosing recommendations, and whether this is associated with better outcomes.
  * Advanced disease is defined as Stage IV (Stage III or IV if multiple myeloma) AND prior chemotherapy in metastatic setting. The PRS is a quantification of eight individual patient risk factors (EORTC guidelines-2010).
  CV: cardiovascular; EORTC: European Organization for Research and Treatment in Cancer; FN: febrile neutropenia; Hb: hemoglobin
Time Frame: as for outcome 1
Population: Evaluable sample
Measure: Number; unit: percentage of participants
Arm/Group | EP2006
Number analyzed (Participants) | 1447
percentage of participants
  Age >=65 years | 41.3
  Advanced disease* | 13.7
  History of FN | 1.9
  No antibiotic prophylaxis | 87.8
  Poor performance and/or nutritional status | 13.1
  Female gender | 61.2
  Hb < 12 g/dL | 39.6
  Renal, CV, or liver disease | 23.1

43. Primary Outcome: Percentage of Patients With Each EORTC-identified Risk Factors for FN in Patients With Chemotherapy Risk 10-20% at Baseline
Description: Objective 3: To determine the extent to which the primary and secondary prophylaxis of FN in cancer patients is in congruence with the EORTC best practice guidelines and dosing recommendations, and whether this is associated with better outcomes.
  * Advanced disease is defined as Stage IV (Stage III or IV if multiple myeloma) AND prior chemotherapy in metastatic setting CV: cardiovascular; EORTC: European Organization for Research and Treatment in Cancer; FN: febrile neutropenia; Hb: hemoglobin
Time Frame: as for outcome 1
Population: Patients with chemotherapy risk 10-20% in evaluable sample
Measure: Number; unit: percentage of patients
Arm/Group | EP2006
Number analyzed (Participants) | 650
percentage of patients
  Age >=65 years | 44.6
  Advanced disease* | 20.8
  History of FN | 2.0
  No antibiotic prophylaxis | 91.3
  Poor performance and/or nutritional status | 13.3
  Female gender | 57.8
  Hb < 12 g/dL | 45.9
  Renal, CV, or liver disease | 26.9

44. Secondary Outcome: Cohort Identification
Description: Objective 7: To identify different latent clusters of end-stage cancer patients receiving chemotherapy and being treated with EP2006 for the treatment or primary or secondary prophylaxis of FN using statistical data-mining techniques to profile patients based on medical history, concomitant comorbid conditions, and current clinical status.
  A two-group solution converged and the groups differentiated on key baseline variables. However, the group sizes were too unevenly distributed for further analysis with the "high risk group" comprised of only 3.0% of the evaluable sample.
  ANC=Absolute Neutrophil Count; CIN=Chemotherapy-Induced Neutropenia; FN=Febrile Neutropenia
Time Frame: as for outcome 1
Population: The evaluable sample consists of all patients who received at least one dose of study medication, had no major protocol violation and have a minimum of enrollment cycle and either one follow-up cycle or study end data with valid outcome data (i.e., ANC or completed CIN/FN data).
Measure: Number; unit: participants
Groups:
- EP2006 - Group 1: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Arm/Group | EP2006 - Group 1
Number analyzed (Participants) | 1447
participants
  EP2006 - Group 1 | 1192
  EP2006 - Group 2 | 43
  Missing | 212

45. Secondary Outcome: Characteristics of Clusters: Hemoglobin Study Start
Description: Objective 7: To identify different latent clusters of end-stage cancer patients receiving chemotherapy and being treated with EP2006 for the treatment or primary or secondary prophylaxis of FN using statistical data-mining techniques to profile patients based on medical history, concomitant comorbid conditions, and current clinical status.
Time Frame: as for outcome 1
Population: A two-group solution converged and the groups differentiated on key baseline variables. However, the group sizes were too unevenly distributed for further analysis with the "high risk group" comprised of only 3.0% of the evaluable sample.
  Only patients with data in each group are analyzed for hemoglobin at study start.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- EP2006 - Group 2: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Arm/Group | EP2006 - Group 1 | EP2006 - Group 2
Number analyzed (Participants) | 1175 | 43
g/dL | 12.35 (1.80) | 11.82 (1.86)

46. Primary Outcome: Patient Risk Score (PRS) for All Patients
Description: Objective 3: To determine the extent to which the primary and secondary prophylaxis of FN in cancer patients is in congruence with the EORTC best practice guidelines and dosing recommendations, and whether this is associated with better outcomes.
  Patient risk score (PRS) shows the individual patient risk for FN.The PRS is a sum of eight weighted individual patient risk factors for FN and results in a possible score of 0 to 11 (highest risk for FN). The risk factors were assigned weights based on the level of risk specified by guidelines and SC consensus (age > 65 years: 3.0; advanced disease: 1.5; history of FN: 3.0; No antibiotic prophylaxis: 0.5; poor performance/nutritional status: 1.5; female gender: 0.5; Hb<12g/dL: 0.5; Renal, CV or liver disease: 0.5).
  Advanced disease: Stage IV or Stage III + prior chemotherapy in metastatic setting; CV: cardiovascular; EORTC: European Organization for Research and Treatment in Cancer; FN: febrile neutropenia
Time Frame: as for outcome 1
Population: Evaluable sample
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EP2006
Number analyzed (Participants) | 1447
Scores on a scale | 2.9 (2.0)

47. Primary Outcome: Patient Risk Score (PRS) for Patients Receiving Chemotherapy With 10-20% FN Risk by Tumor Type
Description: as for outcome 46
Time Frame: as for outcome 1
Population: Patients with chemotherapy with 10-20% risk of FN in the evaluable sample by tumor type
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- EP2006 - All Patients: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN (all patients).
- EP2006 - Solid Tumor: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN (Solid tumor).
- EP2006 - Hematological Tumor: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN (Hematological tumor).
Arm/Group | EP2006 - All Patients | EP2006 - Solid Tumor | EP2006 - Hematological Tumor
Number analyzed (Participants) | 650 | 568 | 82
Scores on a scale | 3.3 (2.0) | 3.2 (1.9) | 3.4 (2.4)

48. Primary Outcome: Percentage of Patients With Each Prophylaxis Decision by Chemotherapy-associated FN Risk
Description: Objective 3: To determine the extent to which the primary and secondary prophylaxis of FN in cancer patients is in congruence with the EORTC best practice guidelines and dosing recommendations, and whether this is associated with better outcomes.
  FN: Febrile Neutropenia; EORTC: European Organisation for Research and Treatment of Cancer
Time Frame: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- EP2006, >20% Chemo-associated FN Risk: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN (>20% chemo-associated FN risk)
- EP2006, 10-20% Chemo-associated FN Risk: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN (10-20% chemo-associated FN risk).
- EP2006, <10% Chemo-associated FN Risk: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN (<10% chemo-associated FN risk).
Arm/Group | EP2006, >20% Chemo-associated FN Risk | EP2006, 10-20% Chemo-associated FN Risk | EP2006, <10% Chemo-associated FN Risk
Number analyzed (Participants) | 640 | 650 | 154
percentage of participants
  Primary prophylaxis: Correctly treated (%) | 35.0 | 17.3 | 0
  Primary prophylaxis:Over-treated (%) | 0 | 13.0 | 6.9
  Secondary prophylaxis: Correctly treated (%) | 0 | 3.1 | 1.2
  Secondary prophylaxis: Under-treated (%) | 9.3 | 8.1 | 0
  Secondary prophylaxis: Over-treated (%) | 0 | 3.5 | 2.6
  Primary prophylaxis: Under-treated (%) | 0 | 0 | 0

49. Primary Outcome: Percentage of Patients With Each Chemotherapy Risk Score (CRS) Result by Tumor Type
Description: Objective 3: To determine the extent to which the primary and secondary prophylaxis of FN in cancer patients is in congruence with the EORTC best practice guidelines and dosing recommendations, and whether this is associated with better outcomes.
  The CRS quantifies whether the decision to initiate EP2006 as either primary or secondary prophylaxis is consistent with the EORTC guideline (2010) recommendation based upon the patient's chemotherapy toxicity (<10%, 10-20% or >20% risk of FN) and the PRS. There are three possible results: under-treated, correctly treated, over-treated
Time Frame: as for outcome 2
Population: Evaluable sample: total and by tumor type
Measure: Number; unit: percentage of patients
Groups:
- EP2006: All Patients: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006: Solid Tumor: Cancer patients (Solid tumor) treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006: Hematological Tumor: Cancer patients (Hematological tumor) treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Arm/Group | EP2006: All Patients | EP2006: Solid Tumor | EP2006: Hematological Tumor
Number analyzed (Participants) | 1444 | 1115 | 329
percentage of patients
  Under-treated (%) | 17.3 | 16.3 | 21.0
  Correctly or Over-treated (%) | 82.5 | 83.7 | 79.0
Statistical Analysis 1: Comparison: EP2006: Solid Tumor vs EP2006: Hematological Tumor; Test type: Superiority or Other; p = 0.2698, Chi-squared; Odds Ratio (OR) = 0.7350, 95% CI 2-sided [0.4255 to 1.2698]

50. Primary Outcome: EP2006 Day of Initiation Relative to Guidelines by Cancer Type
Description: Objective 3: To determine the extent to which the primary and secondary prophylaxis of FN in cancer patients is in congruence with the EORTC best practice guidelines and dosing recommendations, and whether this is associated with better outcomes.
  ^ 168 cycles in which ZARZIO® was initiated on day 4 or later involved regimens deemed by the Study Steering Committee to be suitable for GCSF initiation any day after chemotherapy (day 1 or later), e.g., etoposide; hence, these patients were re-classified as being within guidelines
  DLBCL- Diffuse Large B-Cell Lymphoma. Guidelines refers to EORTC 2010 guidelines
Time Frame: as for outcome 2
Population: Number of cycles with initiation on different days during chemotherapy for evaluable sample. A patient may have initiated EP2006 during chemotherapy on different days for different cycles. The categories therefore are not mutually exclusive on a patient level and the sum of patients may therefore exceed the sample size.
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Groups:
- EP2006: EP2006 Initiation During Chemotherapy (Day 0): Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN (EP2006 initiation during chemotherapy, day 0).
- EP2006: EP 2006 Initiation Per Guidelines (Days 1-3): Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN (EP 2006 initiation per guidelines (days 1-3).
- EP2006: EP2006 Initiation Later (Day 4 or More)^: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN (EP2006 initiation later (day 4 or more).
Arm/Group | EP2006: EP2006 Initiation During Chemotherapy (Day 0) | EP2006: EP 2006 Initiation Per Guidelines (Days 1-3) | EP2006: EP2006 Initiation Later (Day 4 or More)^
Number analyzed (Participants) | 234 | 851 | 473
Number analyzed (cycles) | 795 | 3320 | 1815
cycles
  Breast | 178 | 1410 | 624
  Lung | 305 | 691 | 225
  Lymphoma (DLBCL) | 23 | 386 | 671
  Ovarian | 109 | 332 | 119
  Prostate | 26 | 278 | 95
  Multiple myeloma | 32 | 167 | 37
  Bladder | 122 | 56 | 44
Statistical Analysis 1: Comparison: EP2006: EP2006 Initiation During Chemotherapy (Day 0) vs EP2006: EP 2006 Initiation Per Guidelines (Days 1-3) vs EP2006: EP2006 Initiation Later (Day 4 or More)^; Test type: Superiority or Other; p < 0.0001, Chi-squared

51. Primary Outcome: GCSF Initiation Score (GIS)
Description: Objective 3: To determine the extent to which the primary and secondary prophylaxis of FN in cancer patients is in congruence with the EORTC best practice guidelines and dosing recommendations, and whether this is associated with better outcomes.
  ANC=Absolute Neutrophil Count; GIS Score 0 (EP2006 initiated on day 0 of chemotherapy or on day 10 or later); GIS Score 0.50 (EP2006 initiated on days 7-9 of chemotherapy); GIS Score 0.75 (EP2006 initiated on days 4-6 of chemotherapy); GIS Score 1.00 (EP2006 initiated per EORTC guidelines (2010) on days 1-3 after chemotherapy)
  ANC=Absolute Neutrophil Count; CIN=Chemotherapy-Induced Neutropenia; EORTC=European Organization for Research and Treatment in Cancer; FN=Febrile Neutropenia; GCSF=Granulocyte Colony-Stimulating Factor; GIS=Granulocyte Colony-Stimulating Factor Initiation Score
Time Frame: as for outcome 2
Population: as for outcome 44
Measure: Number; unit: Percent of participants
Arm/Group | EP2006
Number analyzed (Participants) | 1423
Percent of participants
  GIS score 0 (%) | 15.9
  GIS score 0.50 (%) | 11.5
  GIS score 0.75 (%) | 16.6
  GIS score 1.0 (%) | 56.0

52. Primary Outcome: GCSF Persistence Score (GPS)
Description: Objective 3: To determine the extent to which the primary and secondary prophylaxis of FN in cancer patients is in congruence with the EORTC best practice guidelines and dosing recommendations, and whether this is associated with better outcomes.
  The GPS grades persistence based on the number of cycles in the line of chemotherapy in which EP2006 was administered, D, relative to the number of cycles in which it should have been continued, C. Thus, the GPS = D/C and ranges from 0 to 1.0
  ANC=Absolute Neutrophil Count; CIN=Chemotherapy-Induced Neutropenia; EORTC=European Organization for Research and Treatment in Cancer; FN=Febrile Neutropenia; GCSF=Granulocyte Colony-Stimulating Factor
Time Frame: as for outcome 2
Population: Patients in the evaluable sample with a GCSF persistence score (GPS).
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1295
participants
  GPS score 0 | 123
  GPS score 0.33 | 2
  GPS score 0.50 | 3
  GPS score 0.60 | 2
  GPS score 0.67 | 4
  GPS score 0.75 | 1
  GPS score 0.80 | 3
  GPS score 1 | 1157

53. Primary Outcome: GCSF Congruence Score (GCS)
Description: Objective 3: To determine the extent to which the primary and secondary prophylaxis of FN in cancer patients is in congruence with the EORTC best practice guidelines and dosing recommendations, and whether this is associated with better outcomes.
  The GCS is computed at the patient level as an overall grade of how congruent actual GCSF treatment is to recommended treatment. The GCS is computed as follows and scores range from 0 to 3: GCS = Σ(CRS + mean GIS over all cycles + GPS), with higher scores indicating higher congruence.
  CRS: Chemotherapy Risk Score (0 or 1 with 1 best); FN: febrile neutropenia; GCSF: granulocyte colony-stimulating factor; GIS=GCSF Initiation Score (0 to 1 with 1 best); GPS=GCSF persistence score (0 to 1 with 1 best);
Time Frame: as for outcome 2
Population: Evaluable sample with GCSF congruence score by tumor type
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- EP2006 - All Patients: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006 - Solid Tumor: Cancer patients (Solid tumor) treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006 - Hematological Tumor: Cancer patients (Hematological tumor) treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Arm/Group | EP2006 - All Patients | EP2006 - Solid Tumor | EP2006 - Hematological Tumor
Number analyzed (Participants) | 1278 | 1015 | 263
scores on a scale | 2.5 (0.6) | 2.5 (0.6) | 2.5 (0.5)

54. Primary Outcome: Absolute Neutrophil Count (ANC) at EP2006 Initiation
Description: Objective 4: To describe hematological outcomes observed in association with primary and secondary prophylactic use of EP2006 in patients at risk for FN; including break-through episodes of FN.
Time Frame: as for outcome 1
Population: Number of patients in evaluable sample with initial ANC result
Measure: Mean (Standard Deviation); unit: Per mm^3
Arm/Group | EP2006
Number analyzed (Participants) | 1283
Per mm^3 | 4429.7 (4725.8)

55. Primary Outcome: Absolute Neutrophil Count (ANC) Across All Cycles
Description: as for outcome 54
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: Per mm^3
Units Other Than Participants: cycles
Groups:
- EP2006 Cycles: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Arm/Group | EP2006 Cycles
Number analyzed (Participants) | 1447
Number analyzed (cycles) | 7792
Per mm^3 | 4585.6 (3889.8)

56. Primary Outcome: Number of Patients With CIN/FN Episodes: Patient Level
Description: Objective 4: To describe hematological outcomes observed in association with primary and secondary prophylactic use of EP2006 in patients at risk for FN; including break-through episodes of FN.
  CIN: Chemotherapy-Induced Neutropenia; FN: Febrile Neutropenia; Chemotherapy disturbance=dose reduction, delay, and/or cancellation; Composite (any of CIN grade 4, FN, CIN/FN-related hospitalization or CIN/FN-related chemotherapy disturbance)
  A patient may fall into more than one or none of the categories displayed.
Time Frame: as for outcome 2
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1447
participants
  CIN any grade | 504
  CIN grade 3/4 | 332
  CIN grade 4 | 191
  FN | 86
  CIN/FN-related hospitalization | 88
  CIN/FN-related chemotherapy disturbance | 138
  Composite | 323

57. Primary Outcome: CIN/FN Episodes: Cycle Level
Description: Objective 4: To describe hematological outcomes observed in association with primary and secondary prophylactic use of EP2006 in patients at risk for FN; including break-through episodes of FN.
  Chemotherapy-Induced Neutropenia (CIN); Febrile Neutropenia (FN); Chemotherapy disturbance=dose reduction, delay, and/or cancellation; Composite (any of CIN grade 4, FN, CIN/FN-related hospitalization [RH] or CIN/FN-related chemotherapy disturbance [RCD])
Time Frame: as for outcome 2
Population: Number of cycles in evaluable sample
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Groups:
- EP2006 Cycle Level: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Arm/Group | EP2006 Cycle Level
Number analyzed (Participants) | 1447
Number analyzed (cycles) | 7570
cycles
  CIN any grade (n=7557) | 1083
  CIN grade 3/4 (n=7541) | 602
  CIN grade 4 (n=7541) | 294
  FN (n=7532) | 105
  CIN/FN-RH (n=7531) | 111
  CIN/FN-RCD (n=6213) | 174
  Composite (n=7570) | 507

58. Primary Outcome: Incidence of Outcomes by Chemotherapy Risk: Patient Level
Description: Objective 5: To describe the distribution of chemotherapy dose delays and reductions, surgery delays and cancellations, radiotherapy delays, dose reductions, and cancellations, and mortality (GCSF-related; FN-related; cancer-related; not related to GCSF, FN, or cancer; all-cause); and estimate the time-to-event for such events over the course of EP2006 treatment.
  Table presents incidences of different outcomes and composite outcome by chemotherapy risk group. ^Composite endpoint includes any of CIN grade 4, FN, CIN/FN-related hospitalization and CIN/FN-related chemotherapy disturbance.
  CIN: Chemotherapy-Induced Neutropenia; FN: Febrile Neutropenia; ANC: Absolute Neutrophil count; GIS: GCSF Initiation Score; Prophylaxis decision mentioned below are relative to EORTC guidelines (2010).
Time Frame: as for outcome 2
Population: Evaluable sample by chemotherapy risk
Measure: Number; unit: percentage of participants
Groups:
- EP2006: Low (<10%) Risk: Cancer patients treated with chemotherapy with low risk(<10%) and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006: Medium (10-20%) Risk: Cancer patients treated with chemotherapy with medium risk(10-20%) and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006: High (>20%) Risk: Cancer patients treated with chemotherapy with high risk(>20%) and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Arm/Group | EP2006: Low (<10%) Risk | EP2006: Medium (10-20%) Risk | EP2006: High (>20%) Risk
Number analyzed (Participants) | 154 | 650 | 640
percentage of participants
  CIN grade 4 | 7.8 | 11.8 | 15.9
  FN | 3.9 | 3.5 | 8.9
  Composite^ | 16.9 | 20.9 | 25.2

59. Primary Outcome: Incidence of CIN/FN-related Chemotherapy Disturbance by EP2006 Prophylaxis Type: Patient Level
Description: Objective 5: To describe the distribution of chemotherapy dose delays and reductions, surgery delays and cancellations, radiotherapy delays, dose reductions, and cancellations, and mortality (GCSF-related; FN-related; cancer-related; not related to GCSF, FN, or cancer; all-cause); and estimate the time-to-event for such events over the course of EP2006 treatment.
  CIN: Chemotherapy-Induced Neutropenia; FN: Febrile Neutropenia; ANC: Absolute Neutrophil count; GIS: GCSF Initiation Score; Prophylaxis decision mentioned below are relative to EORTC guidelines (2010).
Time Frame: as for outcome 2
Population: Evaluable sample by prophylaxis type
Measure: Number; unit: Percentage of participants
Arm/Group | EP2006: Primary Prophylaxis | EP2006: Secondary Prophylaxis
Number analyzed (Participants) | 1046 | 401
Percentage of participants | 7.5 | 15.0

60. Primary Outcome: Incidence of CIN/FN-related Hospitalization Outcomes by EP2006 Practice Patterns (Relative to Guidelines): Patient Level
Description: Objective 5: To describe the distribution of chemotherapy dose delays and reductions, surgery delays and cancellations, radiotherapy delays, dose reductions, and cancellations, and mortality (GCSF-related; FN-related; cancer-related; not related to GCSF, FN, or cancer; all-cause); and estimate the time-to-event for such events over the course of EP2006 treatment.
  Table presents incidences of different outcomes and composite outcome by prophylaxis decision (relative to guidelines). ^Composite endpoint includes any of CIN grade 4, FN, CIN/FN-related hospitalization and CIN/FN-related chemotherapy disturbance.
  CIN: Chemotherapy-Induced Neutropenia; FN: Febrile Neutropenia; ANC: Absolute Neutrophil count; GIS: GCSF Initiation Score; Prophylaxis decision mentioned below are relative to EORTC guidelines (2010).
Time Frame: as for outcome 2
Population: Evaluable sample by prophylaxis decision (relative to guidelines)
Measure: Number; unit: percentage of participants
Groups:
- EP2006: Undertreated: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN, undertreated relative to guidelines
- EP2006: Correctly Treated: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN, correctly treated relative to guidelines
- EP2006: Overtreated: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN, overtreated relative to guidelines.
Arm/Group | EP2006: Undertreated | EP2006: Correctly Treated | EP2006: Overtreated
Number analyzed (Participants) | 251 | 817 | 376
percentage of participants
  CIN grade 4 | 12.0 | 16.8 | 6.4
  FN | 5.2 | 8.0 | 2.1
  CIN/FN-related hospitalization | 8.0 | 7.1 | 2.7
  CIN/FN-related chemotherapy disturbance | 14.7 | 8.8 | 7.7
  Composite^ | 24.7 | 26.0 | 13.0

61. Primary Outcome: Incidence of CIN Grade 4 Episodes by EP2006 Dose: Patient Level
Description: as for outcome 59
Time Frame: as for outcome 2
Population: Evaluable sample by study drug dose
Measure: Number; unit: percentage of participants
Groups:
- EP2006: 30MIU/Day: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN, treated with 30MIU/day
- EP2006: 48MIU/Day: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN, treated with 48MIU/day
Arm/Group | EP2006: 30MIU/Day | EP2006: 48MIU/Day
Number analyzed (Participants) | 815 | 610
percentage of participants | 11.3 | 15.9

62. Primary Outcome: Incidence of Outcomes by Mean GIS: Patient Level
Description: Objective 5: To describe the distribution of chemotherapy dose delays and reductions, surgery delays and cancellations, radiotherapy delays, dose reductions, and cancellations, and mortality (GCSF-related; FN-related; cancer-related; not related to GCSF, FN, or cancer; all-cause); and estimate the time-to-event for such events over the course of EP2006 treatment.
  Table presents incidences of outcomes by day (mean GIS over all visits). ^Composite outcome includes CIN grade 4, FN, CIN/FN-related hospitalization and CIN/FN-related chemotherapy disturbance
  CIN: Chemotherapy-Induced Neutropenia; FN: Febrile Neutropenia; ANC: Absolute Neutrophil count; GIS: GCSF Initiation Score; Prophylaxis decision mentioned below are relative to EORTC guidelines (2010).
Time Frame: as for outcome 2
Population: Evaluable sample by mean GIS
Measure: Number; unit: percentage of participants
Groups:
- EP2006: Mean GIS 0-0.5: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN with mean GIS 0-0.5
- EP2006: Mean GIS 0.51-0.99: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN with mean GIS 0.51-0.99
- EP2006: Mean GIS 1: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN with mean GIS 1
Arm/Group | EP2006: Mean GIS 0-0.5 | EP2006: Mean GIS 0.51-0.99 | EP2006: Mean GIS 1
Number analyzed (Participants) | 390 | 308 | 725
percentage of participants
  CIN grade 4 | 17.7 | 17.5 | 9.2
  Composite^ | 26.9 | 24.7 | 18.9

63. Primary Outcome: Incidence of Outcomes: Cycles Level
Description: Objective 5: To describe the distribution of chemotherapy dose delays and reductions, surgery delays and cancellations, radiotherapy delays, dose reductions, and cancellations, and mortality (GCSF-related; FN-related; cancer-related; not related to GCSF, FN, or cancer; all-cause); and estimate the time-to-event for such events over the course of EP2006 treatment.
  Table presents incidences of outcomes on a cycle level. ^Composite outcome includes CIN grade 4, FN, CIN/FN-related hospitalization and CIN/FN-related chemotherapy disturbance
  CIN: Chemotherapy-Induced Neutropenia; FN: Febrile Neutropenia; ANC: Absolute Neutrophil count; GIS: GCSF Initiation Score; Prophylaxis decision mentioned below are relative to EORTC guidelines (2010).
Time Frame: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | EP2006
Number analyzed (Participants) | 1447
Percentage of participants
  CIN grade 4 | 3.9
  FN | 1.4
  CIN/FN-related hospitalization | 1.5
  CIN/FN-related chemotherapy disturbance | 2.8
  Composite^ | 6.7

64. Primary Outcome: Incidence of Outcomes by Day of Study Drug Initiation: Cycle Level
Description: Objective 5: To describe the distribution of chemotherapy dose delays and reductions, surgery delays and cancellations, radiotherapy delays, dose reductions, and cancellations, and mortality (GCSF-related; FN-related; cancer-related; not related to GCSF, FN, or cancer; all-cause); and estimate the time-to-event for such events over the course of EP2006 treatment.
  Table presents incidences of outcomes on a cycle level by day of study drug initiation. ^Composite outcome includes CIN grade 4, FN, CIN/FN-related hospitalization and CIN/FN-related chemotherapy disturbance
  CIN: Chemotherapy-Induced Neutropenia; FN: Febrile Neutropenia; ANC: Absolute Neutrophil count; GIS: GCSF Initiation Score; Prophylaxis decision mentioned below are relative to EORTC guidelines (2010). *Day of EP2006 initiation- Day 0 (during chemotherapy); **Day of EP2006 initiation- Days 1-3 (per guidelines)
Time Frame: as for outcome 2
Population: Evaluable sample by day of study drug initiation. As these are cycle-level analyses and since patients can be in more than one category over the course of the study, the sum of patients of all three categories may exceed the sample size.
Measure: Number; unit: percentage of participants
Groups:
- EP2006: Day 0 (During Chemotherapy): Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN that initiated study drug on day 0 (during chemotherapy)
- EP2006: Days 1-3 (Per Guidelines): Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN that initiated study drug on days 1-3 (per guidelines)
- EP2006: Day 4 or Later: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN that initiated study drug on day 4 or later
Arm/Group | EP2006: Day 0 (During Chemotherapy) | EP2006: Days 1-3 (Per Guidelines) | EP2006: Day 4 or Later
Number analyzed (Participants) | 234 | 851 | 473
percentage of participants
  CIN grade 4 | 3.1 | 2.8 | 7.3
  FN | 1.0 | 1.2 | 2.1
  Composite^ | 5.8 | 5.4 | 9.1

65. Primary Outcome: Incidence of Outcomes by Study Drug Duration: Cycle Level
Description: Objective 5: To describe the distribution of chemotherapy dose delays and reductions, surgery delays and cancellations, radiotherapy delays, dose reductions, and cancellations, and mortality (GCSF-related; FN-related; cancer-related; not related to GCSF, FN, or cancer; all-cause); and estimate the time-to-event for such events over the course of EP2006 treatment.
  Table presents incidences of outcomes on a cycle level by study drug duration. ^Composite outcome includes CIN grade 4, FN, CIN/FN-related hospitalization and CIN/FN-related chemotherapy disturbance
  CIN: Chemotherapy-Induced Neutropenia; FN: Febrile Neutropenia;
Time Frame: as for outcome 2
Population: Evaluable sample by study drug duration. As these are cycle-level analyses and since patients can be in more than one category over the course of the study, the sum of patients of all three categories may exceed the sample size.
Measure: Number; unit: percentage of participants
Groups:
- EP2006: 1-3 Days Duration: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN with 1-3 days of study drug duration.
- EP2006: 4-5 Days Duration: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN with 4-5 days of study drug duration.
- EP2006: >=6 Days Duration: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN with >=6 days of study drug duration.
Arm/Group | EP2006: 1-3 Days Duration | EP2006: 4-5 Days Duration | EP2006: >=6 Days Duration
Number analyzed (Participants) | 380 | 784 | 419
percentage of participants
  CIN grade 4 | 3.6 | 3.9 | 5.5
  FN | 1.2 | 1.2 | 2.2
  CIN/FN-related chemotherapy disturbance | 2.0 | 2.1 | 4.7
  Composite^ | 6.0 | 5.8 | 9.3

66. Primary Outcome: Number of Patients by Cause of Death
Description: Objective 5: To describe the distribution of chemotherapy dose delays and reductions, surgery delays and cancellations, radiotherapy delays, dose reductions, and cancellations, and mortality (GCSF-related; FN-related; cancer-related; not related to GCSF, FN, or cancer; all-cause); and estimate the time-to-event for such events over the course of EP2006 treatment.
Time Frame: as for outcome 2
Population: Safety population, i.e. all patients who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1496
participants
  All cause | 61
  Cancer-related | 41
  Non-cancer related | 14
  Cause of death specified as "unknown" | 4
  Cause of death not documented | 2

67. Primary Outcome: Number of Participants With All-cause Mortality by Any/no Grade 4 CIN and/or FN
Description: Objective 5: To describe the distribution of chemotherapy dose delays and reductions, surgery delays and cancellations, radiotherapy delays, dose reductions, and cancellations, and mortality (GCSF-related; FN-related; cancer-related; not related to GCSF, FN, or cancer; all-cause); and estimate the time-to-event for such events over the course of EP2006 treatment.
  Table shows number of patients that died in each group.
  CIN: chemotherapy-induced neutropenia; FN: febrile neutropenia
Time Frame: as for outcome 2
Population: Evaluable sample by any/no grade 4 CIN/FN
Measure: Number; unit: participants
Groups:
- EP2006: Any Grade 4 CIN/FN: Cancer patients with any grade 4 CIN/FIN treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006: No Grade 4 CIN/FN: Cancer patients with no grade 4 CIN/FIN treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Arm/Group | EP2006: Any Grade 4 CIN/FN | EP2006: No Grade 4 CIN/FN
Number analyzed (Participants) | 221 | 1226
participants | 10 | 46
Statistical Analysis 1: Comparison: EP2006: Any Grade 4 CIN/FN vs EP2006: No Grade 4 CIN/FN; Test type: Superiority or Other; p = 0.5977, Log Rank

68. Primary Outcome: Number of Participants With All-cause Mortality by CIN/FN-related Chemotherapy Disturbance
Description: Objective 5: To describe the distribution of chemotherapy dose delays and reductions, surgery delays and cancellations, radiotherapy delays, dose reductions, and cancellations, and mortality (GCSF-related; FN-related; cancer-related; not related to GCSF, FN, or cancer; all-cause); and estimate the time-to-event for such events over the course of EP2006 treatment.
  Table shows number of patients who died by any or no CIN/FN related chemotherapy disturbance.
  CIN: chemotherapy-induced neutropenia; FN: febrile neutropenia
Time Frame: as for outcome 2
Population: Evaluable sample by any or no CIN/FN related chemotherapy disturbance.
Measure: Number; unit: participants
Groups:
- EP2006: Any CIN/FN-related Chemotherapy Disturbance: Cancer patients having any CIN/FN-related chemotherapy disturbance treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006: no CIN/FN-related Chemotherapy Disturbance: Cancer patients having no CIN/FN-related chemotherapy disturbance treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Arm/Group | EP2006: Any CIN/FN-related Chemotherapy Disturbance | EP2006: no CIN/FN-related Chemotherapy Disturbance
Number analyzed (Participants) | 138 | 1309
participants | 3 | 53
Statistical Analysis 1: Comparison: EP2006: Any CIN/FN-related Chemotherapy Disturbance vs EP2006: no CIN/FN-related Chemotherapy Disturbance; Test type: Superiority or Other; p = 0.2435, Log Rank

69. Primary Outcome: Number of Participants With Cancer-related Mortality by Any/no Grade 4 CIN or FN
Description: Objective 5: To describe the distribution of chemotherapy dose delays and reductions, surgery delays and cancellations, radiotherapy delays, dose reductions, and cancellations, and mortality (GCSF-related; FN-related; cancer-related; not related to GCSF, FN, or cancer; all-cause); and estimate the time-to-event for such events over the course of EP2006 treatment.
  Table presents number of patients that had a cancer-related death by any/no grade 4 CIN or FN
  CIN: chemotherapy-induced neutropenia; FN: febrile neutropenia
Time Frame: as for outcome 2
Population: Evaluable sample by any/no grade 4 CIN or FN with data
Measure: Number; unit: participants
Groups:
- EP2006: Any Grade 4 CIN/FN: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN with any grade 4 CIN/FN
- EP2006: No Grade 4 CIN/FN: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN with no grade 4 CIN/FN
Arm/Group | EP2006: Any Grade 4 CIN/FN | EP2006: No Grade 4 CIN/FN
Number analyzed (Participants) | 221 | 1220
participants | 6 | 29
Statistical Analysis 1: Comparison: EP2006: Any Grade 4 CIN/FN vs EP2006: No Grade 4 CIN/FN; Test type: Superiority or Other; p = 0.7630, Log Rank

70. Primary Outcome: Number of Participants With Cancer-related Mortality by Any CIN/FN-related Chemotherapy Disturbance
Description: Objective 5: To describe the distribution of chemotherapy dose delays and reductions, surgery delays and cancellations, radiotherapy delays, dose reductions, and cancellations, and mortality (GCSF-related; FN-related; cancer-related; not related to GCSF, FN, or cancer; all-cause); and estimate the time-to-event for such events over the course of EP2006 treatment.
  Table presents number of patients who had a cancer-related death by any/no CIN/FN-related chemotherapy disturbance
  CIN: chemotherapy-induced neutropenia; FN: febrile neutropenia
Time Frame: as for outcome 2
Population: Evaluable sample by any/no CIN/FN-related chemotherapy disturbance with data
Measure: Number; unit: participants
Groups:
- EP2006: Any CIN/FN-related Chemotherapy Disturbance: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN who had any CIN/FN-related chemotherapy disturbance
- EP2006: No CIN/FN-related Chemotherapy Disturbance: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN who had no CIN/FN-related chemotherapy disturbance
Arm/Group | EP2006: Any CIN/FN-related Chemotherapy Disturbance | EP2006: No CIN/FN-related Chemotherapy Disturbance
Number analyzed (Participants) | 138 | 1303
participants | 2 | 33
Statistical Analysis 1: Comparison: EP2006: Any CIN/FN-related Chemotherapy Disturbance vs EP2006: No CIN/FN-related Chemotherapy Disturbance; Test type: Superiority or Other; p = 0.3830, Log Rank

71. Primary Outcome: Number of Participants With Any CIN/FN-related Chemotherapy Disturbance by Prophylaxis Type
Description: Objective 5: To describe the distribution of chemotherapy dose delays and reductions, surgery delays and cancellations, radiotherapy delays, dose reductions, and cancellations, and mortality (GCSF-related; FN-related; cancer-related; not related to GCSF, FN, or cancer; all-cause); and estimate the time-to-event for such events over the course of EP2006 treatment.
  Table presents number of patients with any CIN/FN-related chemotherapy disturbance by prophylaxis type.
  CIN: chemotherapy-induced neutropenia; FN: febrile neutropenia
Time Frame: as for outcome 2
Population: Evaluable sample by prophylaxis type
Measure: Number; unit: participants
Arm/Group | EP2006: Primary Prophylaxis | EP2006: Secondary Prophylaxis
Number analyzed (Participants) | 1046 | 401
participants | 78 | 60
Statistical Analysis 1: Comparison: EP2006: Primary Prophylaxis vs EP2006: Secondary Prophylaxis; Test type: Superiority or Other; p = 0.0002, Log Rank

72. Primary Outcome: Number of Participants With Any CIN/FN-related Chemotherapy Disturbance by Treatment Decision
Description: Objective 5: To describe the distribution of chemotherapy dose delays and reductions, surgery delays and cancellations, radiotherapy delays, dose reductions, and cancellations, and mortality (GCSF-related; FN-related; cancer-related; not related to GCSF, FN, or cancer; all-cause); and estimate the time-to-event for such events over the course of EP2006 treatment.
  Table presents number of patients with any CIN/FN-related chemotherapy disturbances by treatment decision.
  CIN: chemotherapy-induced neutropenia; FN: febrile neutropenia
Time Frame: as for outcome 2
Population: Evaluable sample by treatment decision with data
Measure: Number; unit: participants
Groups:
- EP2006: Undertreated: Undertreated cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006: Correctly Treated: Correctly treated cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
- EP2006: Over Treated: Over treated cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN.
Arm/Group | EP2006: Undertreated | EP2006: Correctly Treated | EP2006: Over Treated
Number analyzed (Participants) | 251 | 817 | 376
participants | 37 | 72 | 29
Statistical Analysis 1: Comparison: EP2006: Undertreated vs EP2006: Correctly Treated vs EP2006: Over Treated; Test type: Superiority or Other; p = 0.0301, Log Rank

73. Primary Outcome: Predictors of Absolute Neutrophil Count
Description: Objective 6: To examine the multilevel determinants (patient, center) of hematological outcomes of primary and secondary prophylaxis with EP2006 to better understand the variability in outcomes achieved.
  Hierarchical modeling was used to test the relationship of patient- and physician/center-level variables and treatment response in terms of ANC. This analysis was conducted at the cycle level using a 1-cycle lag between treatment patterns and outcomes, that is study drug treatment patterns in one cycle predicted the ANC value at the beginning of the next cycle. Log-transformed ANC values were used.
  Table presents predictors for ANC: GCSF decision, study drug dose, tumor type, patient gender, ECOG, Hb
  Since log-transformed Absolute Neutrophil Count (ANC) values were used, Exp(beta) can be interpreted in terms of % change in ANC for each unit change in predictor or for each category relative to the referent (for categorical variables); Hb=Hemoglobin
Time Frame: as for outcome 2
Population: Cycles for patients in evaluable sample with data
Measure: Number; unit: participants
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1185
Number analyzed (cycles) | 4333
participants | 1185
Statistical Analysis 1: Comparison: EP2006; GCSF treatment decision (under vs correct) as predictor for ANC; Test type: Superiority or Other; p = 0.0683, Regression, Logistic; degrees of freedom: 3181; Slope = 0.92, 95% CI 2-sided [0.84 to 1.01]
Statistical Analysis 2: Comparison: EP2006; GCSF decision (Over vs correct) as predictor for ANC; Test type: Superiority or Other; p = 0.0019, Regression, Logistic; degrees of freedom: 3181; Slope = 0.89, 95% CI 2-sided [0.82 to 0.96]
Statistical Analysis 3: Comparison: EP2006; GCSF decision (Under vs over) as predictor for ANC; Test type: Superiority or Other; p = 0.4469, Regression, Logistic; degrees of freedom: 3181; Slope = 1.04, 95% CI 2-sided [0.94 to 1.15]
Statistical Analysis 4: Comparison: EP2006; Study drug dose (higher vs lower) as predictor for ANC; Test type: Superiority or Other; p = 0.0079, Regression, Logistic; Slope = 1.11, 95% CI 2-sided [1.03 to 1.19]
Statistical Analysis 5: Comparison: EP2006; Tumor type (hematological vs solid) as predictor for ANC; Test type: Superiority or Other; p = 0.0004, Regression, Logistic; Slope = 0.81, 95% CI 2-sided [0.72 to 0.91]
Statistical Analysis 6: Comparison: EP2006; Patient gender (female vs male) as predictor for ANC; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Slope = 0.86, 95% CI 2-sided [0.80 to 0.92]
Statistical Analysis 7: Comparison: EP2006; ECOG (per 1 point) as predictor for ANC; Test type: Superiority or Other; p = 0.0235, Regression, Linear; Slope = 1.04, 95% CI 2-sided [1.01 to 1.08]
Statistical Analysis 8: Comparison: EP2006; Hb (per g/dL) as predictor for ANC; Test type: Superiority or Other; p < 0.0001, Regression, Linear; Slope = 1.03, 95% CI 2-sided [1.02 to 1.05]

74. Primary Outcome: Patient/Center-level Covariance Parameter Estimates of Absolute Neutrophil Count
Description: Objective 6: To examine the multilevel determinants (patient, center) of hematological outcomes of primary and secondary prophylaxis with EP2006 to better understand the variability in outcomes achieved.
  Mean and standard error estimated from ANCOVA
Time Frame: as for outcome 2
Population: Evaluable sample
Measure: Number; unit: participants
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1185
Number analyzed (cycles) | 4333
participants | 1185
Statistical Analysis 1: Comparison: EP2006; ANCOVA model was used taking into account center, patient within center-level and within-patient level (over time). This appendix describes the center-level; Test type: Superiority or Other; p = 0.0003, ANCOVA; Intra-class correlation coefficient = 0.09 — The intra-class correlation coefficient (ICC) was computed to quantify the variability in patient outcome attributable to within-center variability before any patient-level determinants are considered
Statistical Analysis 2: Comparison: EP2006; ANCOVA model was used taking into account center, patient within center-level and within-patient level (over time). This appendix describes the patient within center-level; Test type: Superiority or Other; p < 0.0001, ANCOVA; Intra-class correlation coefficient = 0.41
Statistical Analysis 3: Comparison: EP2006; ANCOVA model was used taking into account center, patient within center-level and within-patient level (over time). This appendix describes the within-patient level; Test type: Superiority or Other; p < 0.0001, ANCOVA; Intra-class correlation coefficient = 0.50

75. Secondary Outcome: Characteristics of Clusters: ECOG Performance Status
Description: Objective 7: To identify different latent clusters of end-stage cancer patients receiving chemotherapy and being treated with EP2006 for the treatment or primary or secondary prophylaxis of FN using statistical data-mining techniques to profile patients based on medical history, concomitant comorbid conditions, and current clinical status.
  ECOG score is a severity scale from 0 to 5 (highest) to grade toxicity and is defined as follows: 0=none, 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=lethal. ECOG is described in more detail by Oken et al, Am J Clin Oncol (CCT) 5:649-655, 1982.
  FN=Febrile Neutropenia; ECOG: European Cooperative Oncology Group
Time Frame: as for outcome 1
Population: A two-group solution converged and the groups differentiated on key baseline variables. However, the group sizes were too unevenly distributed for further analysis with the "high risk group" comprised of only 3.0% of the evaluable sample.
  Only patients with data in each group are analyzed for ECOG performance status.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EP2006 - Group 1 | EP2006 - Group 2
Number analyzed (Participants) | 1145 | 39
Scores on a scale | 0.75 (0.72) | 0.87 (0.61)

76. Secondary Outcome: Characteristics of Clusters: Cancer Stage
Description: Objective 7: To identify different latent clusters of end-stage cancer patients receiving chemotherapy and being treated with EP2006 for the treatment or primary or secondary prophylaxis of FN using statistical data-mining techniques to profile patients based on medical history, concomitant comorbid conditions, and current clinical status.
  FN=Febrile Neutropenia
Time Frame: as for outcome 1
Population: A two-group solution converged and the groups differentiated on key baseline variables. However, the group sizes were too unevenly distributed for further analysis with the "high risk group" comprised of only 3.0% of the evaluable sample.
  Only patients with data in each group are analyzed for cancer stage.
Measure: Number; unit: participants
Arm/Group | EP2006 - Group 1 | EP2006 - Group 2
Number analyzed (Participants) | 1192 | 41
participants
  Cancer Stage III | 511 | 12
  Cancer Stage IV | 681 | 29

77. Secondary Outcome: Characteristics of Clusters: History of Antibiotic Use for CIN
Description: Objective 7: To identify different latent clusters of end-stage cancer patients receiving chemotherapy and being treated with EP2006 for the treatment or primary or secondary prophylaxis of FN using statistical data-mining techniques to profile patients based on medical history, concomitant comorbid conditions, and current clinical status.
  CIN=Chemotherapy Induced Neutropenia; FN=Febrile Neutropenia
Time Frame: as for outcome 1
Population: A two-group solution converged and the groups differentiated on key baseline variables. However, the group sizes were too unevenly distributed for further analysis with the "high risk group" comprised of only 3.0% of the evaluable sample.
  Only patients with data in each group are analyzed for history of antibiotic use for CIN.
Measure: Number; unit: participants
Arm/Group | EP2006 - Group 1 | EP2006 - Group 2
Number analyzed (Participants) | 1192 | 41
participants
  No history for antibiotic use for CIN | 1190 | 17
  History for antibiotic use for CIN (Yes) | 2 | 24

78. Secondary Outcome: Characteristics of Clusters: Liver, Renal and/or Cardiovascular Disease
Description: as for outcome 76
Time Frame: as for outcome 1
Population: A two-group solution converged and the groups differentiated on key baseline variables. However, the group sizes were too unevenly distributed for further analysis with the "high risk group" comprised of only 3.0% of the evaluable sample.
  Only patients with data in each group are analyzed for liver, renal and/or cardiovascular disease.
Measure: Number; unit: participants
Arm/Group | EP2006 - Group 1 | EP2006 - Group 2
Number analyzed (Participants) | 1192 | 41
participants
  No Liver, renal and/or cardiovascular disease | 931 | 19
  Liver, renal and/or cardiovascular disease (Yes) | 261 | 22

79. Secondary Outcome: Modeling Grade 4 CIN Episode: Cycle Level
Description: Objective 8: To model patient- and center-level variables between patients who responded and those who did not respond to primary or secondary prophylaxis with EP2006.
  Objective 9: To model patient- and center-level variables between patients who had chemotherapy dose delays or reductions, surgery delays and cancellations, and radiotherapy delays, dose reductions, or cancellations vs. no such events during the course of primary or secondary prophylaxis with EP2006
  Only results with a p-value of <0.05 are added as statistical analyses appendices.
  CI: confidence interval; CIN: chemotherapy-induced neutropenia; GCSF: granulocyte colony-stimulating factor; GIS: GCSF Initiation Score
Time Frame: as for outcome 2
Population: Number of cycles in evaluable sample with any grade 4 CIN data
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1078
Number analyzed (cycles) | 5514
cycles | 294
Statistical Analysis 1: Comparison: EP2006; GIS (1 vs. 0) as cycle-level predictor for CIN grade 4 episode; Test type: Superiority or Other; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 0.544, 95% CI 2-sided [0.365 to 0.812]
Statistical Analysis 2: Comparison: EP2006; Concomitant antibiotic prophylaxis as cycle-level predictor for CIN grade 4 episode; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.795, 95% CI 2-sided [3.242 to 7.092]
Statistical Analysis 3: Comparison: EP2006; CIN1/4 in previous cycle as cycle-level predictor for CIN grade 4 episode; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.083, 95% CI 2-sided [3.242 to 7.092]
Statistical Analysis 4: Comparison: EP2006; History of CIN Grade 4 at enrollment as patient-level predictor for CIN grade 4 episode; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.460, 95% CI 2-sided [1.542 to 3.925]
Statistical Analysis 5: Comparison: EP2006; Over- vs. correctly prophylacted as patient-level predictor for CIN grade 4 episode; Test type: Superiority or Other; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 0.452, 95% CI 2-sided [0.267 to 0.766]

80. Secondary Outcome: Modeling Grade 4 CIN Episode: Patient Level
Description: Objective 8: To model patient- and center-level variables between patients who responded and those who did not respond to primary or secondary prophylaxis with EP2006.
  Objective 9: To model patient- and center-level variables between patients who had chemotherapy dose delays or reductions, surgery delays and cancellations, and radiotherapy delays, dose reductions, or cancellations vs. no such events during the course of primary or secondary prophylaxis with EP2006
  Only results with a p-value of <0.05 are shown in the statistical appendices.
  H/o=History of; CI=confidence interval; CIN=chemotherapy-induced neutropenia
Time Frame: as for outcome 2
Population: Evaluable sample with data
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1323
participants | 191
Statistical Analysis 1: Comparison: EP2006; History of CIN Grade 4 at enrollment as patient-level predictor for CIN grade 4 episode; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 2.925, 95% CI 2-sided [1.592 to 5.374]
Statistical Analysis 2: Comparison: EP2006; Concomitant antibiotic prophylaxis as patient-level predictor for CIN grade 4 episode; Test type: Superiority or Other; p = 0.005, Regression, Logistic; Odds Ratio (OR) = 2.572, 95% CI 2-sided [1.331 to 4.969]
Statistical Analysis 3: Comparison: EP2006; Over- vs. correctly prophylacted as patient-level predictor for CIN grade 4 episode; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.328, 95% CI 2-sided [0.193 to 0.557]

81. Secondary Outcome: Modeling FN Episode: Cycle Level
Description: Objective 8: To model patient- and center-level variables between patients who responded and those who did not respond to primary or secondary prophylaxis with EP2006.
  Objective 9: To model patient- and center-level variables between patients who had chemotherapy dose delays or reductions, surgery delays and cancellations, and radiotherapy delays, dose reductions, or cancellations vs. no such events during the course of primary or secondary prophylaxis with EP2006.
  Only results with a p-value of <0.05 are shown in the statistical appendices.
  CI: confidence interval; CIN: chemotherapy-induced neutropenia; FN: febrile neutropenia; ECOG: Eastern Cooperative Oncology Group
Time Frame: as for outcome 2
Population: Number of cycles of patients in evaluable sample with FN episode data
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1273
Number analyzed (cycles) | 6362
cycles | 105
Statistical Analysis 1: Comparison: EP2006; ECOG score (per 1 point) as cycle-level predictor for FN episode; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.673, 95% CI 2-sided [1.284 to 2.179]
Statistical Analysis 2: Comparison: EP2006; Concomitant antibiotic prophylaxis as cycle-level predictor for FN episode; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.704, 95% CI 2-sided [2.777 to 7.968]
Statistical Analysis 3: Comparison: EP2006; CIN1/4 in previous cycle as cycle-level predictor for FN episode; Test type: Superiority or Other; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 2.190, 95% CI 2-sided [1.342 to 3.574]
Statistical Analysis 4: Comparison: EP2006; History of anaemia at enrollment as patient-level predictor for FN episode; Test type: Superiority or Other; p = 0.010, Regression, Logistic; Odds Ratio (OR) = 0.215, 95% CI 2-sided [0.067 to 0.687]
Statistical Analysis 5: Comparison: EP2006; Under- vs. over-prophylacted as patient-level predictor for FN episode; Test type: Superiority or Other; p = 0.025, Regression, Logistic; Odds Ratio (OR) = 3.501, 95% CI 2-sided [1.169 to 10.487]

82. Secondary Outcome: Modeling FN Episode: Patient Level
Description: Objective 8: To model patient- and center-level variables between patients who responded and those who did not respond to primary or secondary prophylaxis with EP2006.
  Objective 9: To model patient- and center-level variables between patients who had chemotherapy dose delays or reductions, surgery delays and cancellations, and radiotherapy delays, dose reductions, or cancellations vs. no such events during the course of primary or secondary prophylaxis with EP2006
  Only results with a p-value of <0.05 are shown in the statistical appendices.
  CI: confidence interval; CIN: chemotherapy-induced neutropenia; FN: febrile neutropenia
Time Frame: as for outcome 2
Population: Evaluable sample with FN episode data
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1376
participants | 86
Statistical Analysis 1: Comparison: EP2006; Patient age (per 1 year) as patient-level predictor for FN episode; Test type: Superiority or Other; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 0.975, 95% CI 2-sided [0.958 to 0.991]
Statistical Analysis 2: Comparison: EP2006; ECOG ≥2 during study as patient-level predictor for FN episode; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.398, 95% CI 2-sided [1.610 to 3.570]
Statistical Analysis 3: Comparison: EP2006; Concomitant antibiotic prophylaxis as patient-level predictor for FN episode; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 2.562, 95% CI 2-sided [1.450 to 4.527]
Statistical Analysis 4: Comparison: EP2006; Over- vs. correctly prophylacted as patient-level predictor for FN episode; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.232, 95% CI 2-sided [0.108 to 0.499]
Statistical Analysis 5: Comparison: EP2006; Under- vs. over-prophylacted as patient-level predictor for FN episode; Test type: Superiority or Other; p = 0.011, Regression, Logistic; Odds Ratio (OR) = 3.261, 95% CI 2-sided [1.315 to 8.084]

83. Secondary Outcome: Modeling CIN/FN-related Hospitalization: Cycle Level
Description: as for outcome 81
Time Frame: as for outcome 2
Population: Number of cycles of patients in evaluable sample with CIN/FN-related hospitalization data
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1383
Number analyzed (cycles) | 6928
cycles | 111
Statistical Analysis 1: Comparison: EP2006; ECOG score (per 1 point) as cycle-level predictor for CIN/FN-related hospitalization; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.814, 95% CI 2-sided [1.397 to 2.355]
Statistical Analysis 2: Comparison: EP2006; Concomitant antibiotic prophylaxis as cycle-level predictor for CIN/FN-related hospitalization; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.296, 95% CI 2-sided [1.791 to 6.065]
Statistical Analysis 3: Comparison: EP2006; CIN1/4 in previous cycles as cycle-level predictor for CIN/FN-related hospitalization; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 2.205, 95% CI 2-sided [1.380 to 3.524]
Statistical Analysis 4: Comparison: EP2006; Under- vs. correctly prophylacted as patient-level predictor for CIN/FN-related hospitalization; Test type: Superiority or Other; p = 0.032, Regression, Logistic; Odds Ratio (OR) = 1.863, 95% CI 2-sided [1.054 to 3.293]
Statistical Analysis 5: Comparison: EP2006; Over- vs. correctly prophylacted as patient-level predictor for CIN/FN-related hospitalization; Test type: Superiority or Other; p = 0.024, Regression, Logistic; Odds Ratio (OR) = 0.385, 95% CI 2-sided [0.168 to 0.879]
Statistical Analysis 6: Comparison: EP2006; Under- vs. over-prophylacted as patient-level predictor for CIN/FN-related hospitalization; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 4.843, 95% CI 2-sided [1.964 to 11.942]

84. Secondary Outcome: Modeling CIN/FN-related Hospitalization: Patient Level
Description: as for outcome 81
Time Frame: as for outcome 2
Population: Evaluable sample with CIN/FN-related hospitalization data
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1387
participants | 88
Statistical Analysis 1: Comparison: EP2006; ECOG ≥2 during study as patient-level predictor for CIN/FN-related hospitalization; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.473, 95% CI 2-sided [1.550 to 3.946]
Statistical Analysis 2: Comparison: EP2006; Over- vs. correctly prophylacted as patient-level predictor for CIN/FN-related hospitalization; Test type: Superiority or Other; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 0.382, 95% CI 2-sided [0.210 to 0.695]
Statistical Analysis 3: Comparison: EP2006; Under- vs. over-prophylacted as patient-level predictor for CIN/FN-related hospitalization; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 3.108, 95% CI 2-sided [1.560 to 6.192]

85. Secondary Outcome: Modeling CIN/FN-related Chemotherapy Disturbance: Cycle Level
Description: Objective 8: To model patient- and center-level variables between patients who responded and those who did not respond to primary or secondary prophylaxis with EP2006.
  Objective 9: To model patient- and center-level variables between patients who had chemotherapy dose delays or reductions, surgery delays and cancellations, and radiotherapy delays, dose reductions, or cancellations vs. no such events during the course of primary or secondary prophylaxis with EP2006.
  Only results with a p-value of <0.05 are shown in the statistical appendices.
  CI: confidence interval; CIN: chemotherapy-induced neutropenia; GCSF: granulocyte colony-stimulating factor; GIS: GCSF Initiation Score; Chemotherapy disturbance=dose reduction, delay, and/or cancellation
Time Frame: as for outcome 2
Population: Cycles of patients in evaluable sample with CIN/FN-related chemotherapy disturbance with data
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1045
Number analyzed (cycles) | 3376
cycles | 174
Statistical Analysis 1: Comparison: EP2006; CIN1/4 in previous cycle as cycle-level predictor for CIN/FN-related chemotherapy disturbance; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 8.931, 95% CI 2-sided [5.426 to 14.699]
Statistical Analysis 2: Comparison: EP2006; Hematological cancer (vs. oncologic) as patient-level predictor for CIN/FN-related chemotherapy disturbance; Test type: Superiority or Other; p = 0.007, Regression, Logistic; Odds Ratio (OR) = 0.336, 95% CI 2-sided [0.152 to 0.740]
Statistical Analysis 3: Comparison: EP2006; Cancer patients seen in 2009 (per 1 patient) as center-level predictor for CIN/FN-related chemotherapy disturbance; Test type: Superiority or Other; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 0.999, 95% CI 2-sided [0.999 to 1.000]
Statistical Analysis 4: Comparison: EP2006; Chemotherapy-treated cancer patients in 2009 (per 1 patient) as center-level predictor for CIN/FN-related chemotherapy disturbance; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.001, 95% CI 2-sided [1.000 to 1.001]
Statistical Analysis 5: Comparison: EP2006; Center type: academic vs non-academic as center-level predictor for CIN/FN-related chemotherapy disturbance; Test type: Superiority or Other; p = 0.024, Regression, Logistic; Odds Ratio (OR) = 2.456, 95% CI 2-sided [1.127 to 5.353]
Statistical Analysis 6: Comparison: EP2006; Center type: academic-affiliated vs non-academic as center-level predictor for CIN/FN-related chemotherapy disturbance; Test type: Superiority or Other; p = 0.010, Regression, Logistic; Odds Ratio (OR) = 3.344, 95% CI 2-sided [1.342 to 8.331]

86. Secondary Outcome: Modeling CIN/FN-related Chemotherapy Disturbance: Patient Level (Patient-level Predictors)
Description: Objective 8: To model patient- and center-level variables between patients who responded and those who did not respond to primary or secondary prophylaxis with EP2006.
  Objective 9: To model patient- and center-level variables between patients who had chemotherapy dose delays or reductions, surgery delays and cancellations, and radiotherapy delays, dose reductions, or cancellations vs. no such events during the course of primary or secondary prophylaxis with EP2006.
  Only results with a p-value of <0.05 are shown in the statistical appendices.
  CI: confidence interval; CIN: chemotherapy-induced neutropenia; FN: febrile neutropenia
Time Frame: as for outcome 2
Population: Evaluable sample with CIN/FN-related chemotherapy disturbance data
Measure: Number; unit: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1334
cycles | 138
Statistical Analysis 1: Comparison: EP2006; Female gender as patient-level predictor for CIN/FN-related chemotherapy disturbance; Test type: Superiority or Other; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 1.965, 95% CI 2-sided [1.218 to 3.172]
Statistical Analysis 2: Comparison: EP2006; History of CIN4 at enrollment as patient-level predictor for CIN/FN-related chemotherapy disturbance; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 2.594, 95% CI 2-sided [1.469 to 4.581]

87. Secondary Outcome: Modeling Composite Outcome (Any of CIN Grade 4, FN, CIN/FN-related Hospitalization, CIN/FN-related Chemotherapy Disturbance): Cycle Level
Description: Objective 8: To model patient- and center-level variables between patients who responded and those who did not respond to primary or secondary prophylaxis with EP2006.
  Objective 9: To model patient- and center-level variables between patients who had chemotherapy dose delays or reductions, surgery delays and cancellations, and radiotherapy delays, dose reductions, or cancellations vs. no such events during the course of primary or secondary prophylaxis with EP2006.
  Only results with a p-value of <0.05 are shown in the statistical appendices.
  CI: confidence interval; CIN: chemotherapy-induced neutropenia; ECOG: Eastern Cooperative Oncology Group; FN: febrile neutropenia; GCSF: granulocyte colony-stimulating factor; GIS: GCSF Initiation Score.
Time Frame: as for outcome 2
Population: Cycles of patients from evaluable sample with composite outcome data
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1529
Number analyzed (cycles) | 5193
cycles | 507
Statistical Analysis 1: Comparison: EP2006; GIS (1 vs. 0) as cycle-level predictor for composite outcome (any of CIN Grade 4, FN, CIN/FN-related hospitalization, CIN/FN-related chemotherapy disturbance); Test type: Superiority or Other; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 0.590, 95% CI 2-sided [0.424 to 0.821]
Statistical Analysis 2: Comparison: EP2006; Zarzio duration: 4-5 days vs. 6 or more as cycle-level predictor for composite outcome (any of CIN Grade 4, FN, CIN/FN-related hospitalization, CIN/FN-related chemotherapy disturbance); Test type: Superiority or Other; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 0.644, 95% CI 2-sided [0.489 to 0.859]
Statistical Analysis 3: Comparison: EP2006; Zarzio duration: 1-3 days vs. 6 or more as cycle-level predictor for composite outcome (any of CIN Grade 4, FN, CIN/FN-related hospitalization, CIN/FN-related chemotherapy disturbance); Test type: Superiority or Other; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 0.579, 95% CI 2-sided [0.398 to 0.842]
Statistical Analysis 4: Comparison: EP2006; ECOG score (per 1 point) as cycle-level predictor for composite outcome (any of CIN Grade 4, FN, CIN/FN-related hospitalization, CIN/FN-related chemotherapy disturbance); Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 1.369, 95% CI 2-sided [1.140 to 1.643]
Statistical Analysis 5: Comparison: EP2006; Concomitant antibiotic prophylaxis as cycle-level predictor for composite outcome (any of CIN Grade 4, FN, CIN/FN-related hospitalization, CIN/FN-related chemotherapy disturbance); Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.499, 95% CI 2-sided [2.456 to 4.985]
Statistical Analysis 6: Comparison: EP2006; CIN1/4 in previous cycle as cycle-level predictor for composite outcome (any of CIN Grade 4, FN, CIN/FN-related hospitalization, CIN/FN-related chemotherapy disturbance); Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.064, 95% CI 2-sided [3.096 to 5.336]
Statistical Analysis 7: Comparison: EP2006; Female gender as patient-level predictor for composite outcome (any of CIN Grade 4, FN, CIN/FN-related hospitalization, CIN/FN-related chemotherapy disturbance); Test type: Superiority or Other; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 1.545, 95% CI 2-sided [1.175 to 2.033]
Statistical Analysis 8: Comparison: EP2006; History of CIN Grade 4 at enrollment as patient-level predictor for composite outcome (any of CIN Grade 4, FN, CIN/FN-related hospitalization, CIN/FN-related chemotherapy disturbance); Test type: Superiority or Other; p = 0.017, Regression, Logistic; Odds Ratio (OR) = 1.596, 95% CI 2-sided [1.088 to 2.340]

88. Secondary Outcome: Modeling Composite Outcome (Any of CIN Grade 4, FN, CIN/FN-related Hospitalization, CIN/FN-related Chemotherapy Disturbance): Patient Level
Description: Objective 8: To model patient- and center-level variables between patients who responded and those who did not respond to primary or secondary prophylaxis with EP2006.
  Objective 9: To model patient- and center-level variables between patients who had chemotherapy dose delays or reductions, surgery delays and cancellations, and radiotherapy delays, dose reductions, or cancellations vs. no such events during the course of primary or secondary prophylaxis with EP2006.
  Only results with a p-value of <0.05 are shown in the statistical appendices.
  CI: confidence interval; CIN: chemotherapy-induced neutropenia; ECOG: Eastern Cooperative Oncology Group; FN: febrile neutropenia; GCSF: granulocyte colony-stimulating factor; GIS: GCSF Initiation Score. H/o repeated infections refers at enrollment; H/o: History of
Time Frame: as for outcome 2
Population: Patients in evaluable sample with composite outcome data
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1291
participants | 323
Statistical Analysis 1: Comparison: EP2006; [analysis description as in outcome 87, analysis 7]; Test type: Superiority or Other; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 1.621, 95% CI 2-sided [1.152 to 2.281]
Statistical Analysis 2: Comparison: EP2006; History of CIN4 at enrollment as patient-level predictor for composite outcome (any of CIN Grade 4, FN, CIN/FN-related hospitalization, CIN/FN-related chemotherapy disturbance); Test type: Superiority or Other; p = 0.005, Regression, Logistic; Odds Ratio (OR) = 1.898, 95% CI 2-sided [1.209 to 2.979]
Statistical Analysis 3: Comparison: EP2006; History of repeated infections at enrollment as patient-level predictor for composite outcome (any of CIN Grade 4, FN, CIN/FN-related hospitalization, CIN/FN-related chemotherapy disturbance); Test type: Superiority or Other; p = 0.016, Regression, Logistic; Odds Ratio (OR) = 2.680, 95% CI 2-sided [1.200 to 5.984]
Statistical Analysis 4: Comparison: EP2006; Over- vs. correctly prophylacted as patient-level predictor for composite outcome (any of CIN Grade 4, FN, CIN/FN-related hospitalization, CIN/FN-related chemotherapy disturbance); Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.438, 95% CI 2-sided [0.291 to 0.660]
Statistical Analysis 5: Comparison: EP2006; Under- vs. over-prophylacted as patient-level predictor for composite outcome (any of CIN Grade 4, FN, CIN/FN-related hospitalization, CIN/FN-related chemotherapy disturbance); Test type: Superiority or Other; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 2.053, 95% CI 2-sided [1.295 to 3.256]
Statistical Analysis 6: Comparison: EP2006; GIS at enrollment (1 vs. 0) as patient-level predictor for composite outcome (any of CIN Grade 4, FN, CIN/FN-related hospitalization, CIN/FN-related chemotherapy disturbance); Test type: Superiority or Other; p = 0.028, Regression, Logistic; Odds Ratio (OR) = 0.558, 95% CI 2-sided [0.332 to 0.939]

89. Secondary Outcome: Patient-level Predictors for All-cause Mortality
Description: Objective 10: To model patient- and center-level variables between patients who died vs. survived during the course of primary or secondary prophylaxis with EP2006, in all patients and those with break-through FN episodes.
  Table presents patient-level predictors for all-cause mortality: history of anemia at enrollment, liver/renal/cardiac comorbidity, poor performance (ECOG >=2) during study
Time Frame: as for outcome 2
Population: Evaluable sample with data
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1272
participants | 1272
Statistical Analysis 1: Comparison: EP2006; Patient level predictor: History of anemia at enrollment; Test type: Superiority or Other; p = 0.0116, Regression, Logistic; Odds Ratio (OR) = 2.2064, 95% CI 2-sided [1.1931 to 4.0803]
Statistical Analysis 2: Comparison: EP2006; Liver/renal/cardiac comorbidity as patient level predictor; Test type: Superiority or Other; p = 0.0057, Regression, Logistic; Odds Ratio (OR) = 2.3049, 95% CI 2-sided [1.2754 to 4.1656]
Statistical Analysis 3: Comparison: EP2006; Poor performance (ECOG >=2) during study as patient level predictor; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 17.5350, 95% CI 2-sided [8.2159 to 37.4243]

90. Primary Outcome: EP2006 Day of Initiation: Cycle Distribution
Description: Objective 2: To describe EP2006 primary or secondary prophylaxis patterns for FN over up to 6 cycles of chemotherapy, with or without prior, concurrent, or later radiotherapy or surgery.
  Table presents number of cycles by day after chemotherapy.
Time Frame: as for outcome 2
Population: Cycles of patients in evaluable sample with day of study drug initiation
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1447
Number analyzed (cycles) | 5930
cycles
  day 0 | 795
  day1 | 1818
  day 2 | 793
  day 3 | 541
  day 4 | 270
  day 5 | 404
  day 6 | 400
  day 7 | 429
  day 8 | 231
  day 9 | 59
  day10 | 49
  day11 | 36
  ≥day12 | 105

91. Primary Outcome: EP2006 Cycles by Treatment Duration
Description: as for outcome 5
Time Frame: as for outcome 2
Population: All cycles from patients in the evaluable sample with study drug duration
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Arm/Group | EP2006
Number analyzed (Participants) | 1447
Number analyzed (cycles) | 5942
cycles
  1 day | 211
  2 days | 339
  3 days | 729
  4 days | 422
  5 days | 2718
  6 days | 385
  7 days | 682
  8 days | 115
  9 days | 53
  10 days | 120
  11 days | 13
  12 days | 20
  13 days | 8
  14 days | 105
  >=15 days | 22

92. Primary Outcome: Incidence of Outcomes
Description: as for outcome 58
Time Frame: as for outcome 2
Population: Evaluable sample
Measure: Number; unit: percentage of participants
Arm/Group | EP2006
Number analyzed (Participants) | 1447
percentage of participants
  CIN grade 4 | 13.2
  FN | 5.9
  CIN/FN related Hospitalization | 6.1
  CIN/FN-related chemotherapy disturbance | 9.5
  Composite^ | 22.3

93. Secondary Outcome: Patient-level Predictor for Cancer-related Mortality
Description: Objective 10: To model patient- and center-level variables between patients who died vs. survived during the course of primary or secondary prophylaxis with EP2006 in all patients and those with break-through FN episodes.
  Table presents patient level predictors for cancer-related mortality: female gender, poor performance (ECOG >=2) during study.
  ECOG score is a severity scale from 0 to 5 (highest) to grade toxicity and is defined as follows: 0=none, 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=lethal. ECOG is described in more detail by Oken et al, Am J Clin Oncol (CCT) 5:649-655, 1982.
Time Frame: as for outcome 2
Population: Evaluable sample with data
Measure: Number; unit: participants
Arm/Group | EP2006
Number analyzed (Participants) | 1385
participants | 1385
Statistical Analysis 1: Comparison: EP2006; Female gender as patient-level predictor for cancer-related mortality; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 14.8703, 95% CI 2-sided [5.9567 to 37.1225]
Statistical Analysis 2: Comparison: EP2006; Poor performance (ECOG >=2) during study as patient-level predictor; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 14.8703, 95% CI 2-sided [5.9567 to 37.1225]

ADVERSE EVENTS:
Time Frame: Patients were evaluated at the enrollment cycle and then re-evaluated at each cycle for a maximum total of 6 cycles; however, the scheduling of these evaluations was left to the discretion of the physician, mean duration of study for 105 days
Description: The occurrence of adverse drug reactions (ADRs) not including not-related (S)AEs was sought by non-directive questioning of the patient at each visit during the study. Only Adverse events with a suspected relationship to EP2006 were collected.
Groups:
- EP2006: Cancer patients treated with chemotherapy and who are prescribed commercially available filgrastim biosimilar for primary or secondary prophylaxis for FN. Number 1496 refers to the total number of patients who received at least one dose of study medication EP2006.
Arm/Group | EP2006
Serious Adverse Events (participants affected / at risk) | 4/1496
Other Adverse Events (participants affected / at risk) | 36/1496
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EP2006 (N=1496)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Vulvul abscess (Infections and infestations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EP2006 (N=1496)
Bone pain (Musculoskeletal and connective tissue disorders) | 24 (33)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (21)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor is the sole owner of all data, results and any work summarizing the Study to which this agreement refers, and it should be noted that the Investigator agrees to their publication by Sponsor in any scientific or medical journal chosen by Sponsor. It should be noted that the Investigator may not make any communications or publications relating to the Study which forms the basis of this agreement, without the prior written agreement of the Sponsor.